Official Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of

Obinutuzumab in Combination With Idasanutlin and Venetoclax in Patients With Relapsed or Refractory Follicular Lymphoma and Obinutuzumab or Rituximab in Combination With Idasanutlin and Venetoclax in Patients With Relapsed or Refractory Diffuse Large B-

Cell Lymphoma

NCT Number: NCT03135262

**Document Date:** DAP Version 3: 02-April-2019

# **DATA ANALYSIS PLAN (DAP) MODULE 2**

| Title: | Harmonize | ed Specificat | ions Docum | ent for the Ir | nHarmony st | udies |
|---|---|---|---|---|---|---|
| Protocol numbers: | BO29561,<br>BH39147 | BO29562, | BO29563, | GO29833, | GO29834, | ВН29812, |
| Author: | | | | | | |
| , Study Statistician & | | | | Date | | |
| Approver: | | | | | | |
| | * | | | Date | | |

<sup>\*</sup> The approver has ensured that key team members have been involved, contributed and reviewed the content of the List of Planned Outputs as described in the DAP Module 2 guideline.

| | | TABLE OF CONTENTS | Page |
|---|---|---|---|
| 1 | INTRODU | JCTION | 6 |
| 2 | DATA HA | NDLING SPECIFICATIONS | 6 |
| | 2.1 | Datacut | 6 |
| | 2.2 | Treatment Definition | 6 |
| | 2.3 | Patient Allocation to Reporting Periods | 7 |
| | 2.4 | Handling of Missing and Incomplete Data | 10 |
| 3 | SUBGRO | UPS | 11 |
| | 3.1 | ABC/GCB subtypes for DLBCL patients | 11 |
| | 3.2 | BCL-2 subgroups for DLBCL patients | 11 |
| | 3.3 | Double hit subgroup (FISH) for DLBCL patients | 12 |
| | 3.4 | Double positive subgroup (IHC) for DLBCL patients | 12 |
| | 3.5 | IPI / FLIPI | 12 |
| 4 | DEMOGR | APHICS, BASELINE DISEASE CHARACTERISTICS AND PROGNOSTIC MARKERS | 13 |
| | 4.1 | Demographics | 13 |
| | 4.2 | Baseline Disease Characteristics and Prognostic Markers | 13 |
| 5 | EFFICACY | 'ANALYSES | 14 |
| | 5.1 | Analysis of Primary Endpoint | 15 |
| | 5.2 | Analysis of Secondary Endpoints | 15 |
| | 5.3 | Analysis of Exploratory Endpoints | |
| | 5.4 | Interim Analyses | 17 |
| 6 | SAFETY A | NALYSES | 17 |
| | 6.1 | Exposure | 17 |
| | 6.2 | Adverse Events | 18 |
| | 6.3 | Concomitant Medications | 25 |
| | 6.4 | Laboratory Data | 25 |
| 7 | PHARMA | COKINETIC ANALYSES | 29 |
| 8 | PROTOCO | OL DEVIATIONS | 30 |
| 9 | REFEREN | CES | 30 |
| 10 | OUTPUT | TEMPLATE | 30 |
| OUT | PUT TEMP | LATES | 31 |
| | 10.1 | Output 1 Summary of Enrollment by Country and Investigator | 31 |
| | 10.2 | Output 2 Patient Disposition | 32 |
| | 10.3 | Output 3 Analysis Populations | 33 |

| 10.4 | Output 4 Listing of Patients Excluded from Analysis Populations | 33 |
|---|---|---|
| 10.5 | Output 5 Summary of Study Drug Completion Status and Reasons of | |
| | Withdrawals from Study Drug | 34 |
| 10.6 | Output 6 Summary of Duration on Treatment and Follow-up | 35 |
| 10.7 | Output 7 Listing of Patients Who Discontinued Early from Study Drug | 36 |
| 10.8 | Output 8 Major Protocol Deviations | 37 |
| 10.9 | Output 9 Listing of Major Protocol Deviations | 38 |
| 10.10 | Output 10 Demographics and Baseline Characteristics | 39 |
| 10.11 | Output 11 Baseline Disease Characteristics and Prognostic Markers | 41 |
| 10.12 | Output 12 Peripheral Neuropathy History | 46 |
| 10.13 | Output 13 Medical History | 47 |
| 10.14 | Output 14 Listing of Previous Systemic Anti-lymphoma Therapy | 48 |
| 10.15 | Output 15 Previous Systemic Anti-lymphoma Therapy | 49 |
| 10.16 | Output 16 Response to Previous Systemic Anti-lymphoma Therapy | 51 |
| 10.17 | Output 17 Listing of Follow-up New Anti-lymphoma Therapy | 52 |
| 10.18 | Output 18 Follow-up New Anti-lymphoma Therapy | 53 |
| 10.19 | Output 19 Concomitant Medication | 54 |
| 10.20 | Output 20 Previous-Concomitant Medications | 55 |
| 10.21 | Output 21 Previous Medications | 55 |
| 10.22 | Output 22 Surgery and Procedure History | 55 |
| 10.23 | Output 23 Glossary of Superclass terms, Preferred Terms and Verbatim | |
| | Terms for Concomitant Medications | 56 |
| 10.24 | Output 24 Listing of Study Drug Exposure | 57 |
| 10.25 | Output 25 Study Drug Exposure during Induction Phase | 58 |
| 10.26 | Output 26 Study Drug Exposure During Maintenance/Consolidation Phase | 59 |
| 10.27 | Output 27 Glossary of Adverse Event Preferred Terms and Investigator- | |
| | Specified Terms | 60 |
| 10.28 | Output 28 Listing of Adverse Events | 61 |
| 10.29 | Output 29 Listing of Serious Adverse Events | 62 |
| 10.30 | Output 30 Listing of Grade 3, 4, 5 Adverse Events | 62 |
| 10.31 | Output 31 Listing of Adverse Events Leading to Discontinuation of Any Stu | |
| | Drug | 62 |
| 10.32 | Output 32 Listing of Adverse Events Leading to Dose Modification or | |
| | Interruption of Any Study Drug | 62 |
| 10.33 | Output 33 Listing of Adverse Events Leading to Death | 62 |
| 10.34 | Output 34 Listing of Adverse Events of Special Interest | |
| 10.35 | Output 35 Listing of Selected Adverse Events | |
| 10.36 | Output 36 Safety Summary | 64 |
| 10.37 | Output 37 Adverse Events | 65 |
| 10.38 | Output 38 Grade 3, 4, 5 Adverse Events | |
| 10.39 | Output 39 Serious Adverse Events | |
| 10.40 | Output 40 Adverse Events Leading to Discontinuation of Any Study Drug | |
| 10.41 | Output 41 Adverse Events of Special Interest | |
| 10.42 | Output 42 Selected Adverse Events | |
| 10.43 | Output 43 Categorical Summary of Adverse Events of Special Interest | 68 |

| 10.44 | Output 44 Categorical Summary of Selected Adverse Events | 69 |
|---|---|---|
| 10.45 | Output 45 Adverse Events by Cycle | 69 |
| 10.46 | Output 46 AE Special Interest by Cycle | 69 |
| 10.47 | Output 47 Selected AE by Cycle | 70 |
| 10.48 | Output 48 Adverse Events by Highest NCI CTCAE Grade | 70 |
| 10.49 | Output 49 Most Common Adverse Event with Incidence $\geqslant$ 5% by Preferr | ed |
| | Term | 72 |
| 10.50 | Output 50 Most Common Grade 3, 4, 5 Adverse Event with Incidence $\geq$ 5 | 5% |
| | by Preferred Term | 72 |
| 10.51 | Output 51 Duration from First Study Treatment Date to Onset of Peripher | ral |
| | Neuropathy | 73 |
| 10.52 | Output 52 Listing of Deaths | 74 |
| 10.53 | Output 53 Deaths | 75 |
| 10.54 | Output 54 Laboratory Test Results Shift Table – Highest NCI CTCAE Grade | e |
| | Post-Baseline | 76 |
| 10.55 | Output 55 Neutrophil Count Recovery | 77 |
| 10.56 | Output 56 Vital Signs Change from Baseline by Visit | 78 |
| 10.57 | Output 57 ECG Results Shift Table | 79 |
| 10.58 | Output 58 Listing of Time-to-Event Endpoints | 81 |
| 10.59 | Output 59 Listing of Tumor Response Assessment | 82 |
| 10.60 | Output 60 CR Rate at End of Induction | 83 |
| 10.61 | Output 61 OR Rate at End of Induction | 85 |
| 10.62 | Output 62 CR Rate at 12 Months after Initiation of Induction | 87 |
| 10.63 | Output 63 Best Overall Response Rate | 88 |
| 10.64 | Output 64 Concordance Analysis Between the IRC Determined and the | |
| | Investigator Determined CR Status | 89 |
| 10.65 | Output 65 Duration of Response | 90 |
| 10.66 | Output 66 Kaplan-Meier Curve of Duration of Response | 91 |
| 10.67 | Output 67 Waterfall Plot of Best Change from Baseline (%) in Indicator | |
| | Lesion Size | 92 |
| 10.68 | Output 68 Spider Plot of Change from Baseline (%) in Indicator Lesion Siz | e |
| | over Time | |
| 10.69 | Output 69 Swimmer Plot of Time to Response and Duration of Response | |
| 10.70 | Output 70 Progression-Free Survival | |
| 10.71 | Output 71 Kaplan-Meier Curve of Progression-free Survival | 96 |
| 10.72 | Output 72 Event-Free Survival | |
| 10.73 | Output 73 Kaplan-Meier Curve of Event-Fee Survival | 97 |
| 10.74 | Output 74 Disease-Free Survival | |
| 10.75 | Output 75 Kaplan-Meier Curve of Disease-Fee Survival | |
| 10.76 | Output 76 Summary of Overall Survival | 98 |
| 10.77 | Output 77 Kaplan-Meier Curve of Overall Survival | 98 |

| | LIST OF APPENDICES | Page |
|---------------|--------------------|------|
| Appendix 1 | Region Categories | 99 |
| DAP M 2 UPDAT | TE LOG | 100 |

#### 1 Introduction

The purpose of this document is to define the specifications required for the analyses and output production for the InHarmony studies (BO29561, BO29562, BO29563, GO29833, GO29834, BH29812). This document should be referred to alongside the harmonized List of Planned Outputs (LoPO) spreadsheet.

## 2 Data Handling Specifications

#### 2.1 Datacut

For primary CSR analyses, each study will have data cut based on the 'clinical cutoff date' (CCOD). Data collected on or before the CCOD will be included in.

For the datacut rules refer to the instructions for 'fixed-cutoff datacut' type on the Global Data Standards Repository (GDSR) Browser - Rules and Definitions for Analysis Data Cuts.

#### 2.2 Treatment Definition

"Chemotherapy" (CT) is defined as at least one dose > 0 of Doxorubicin, Bendamustine, Cyclophosphamide, Vincristine or Prednisone/Prednisolone/Methylprednisolone (=steroids). Steroids are only counted as part of Chemotherapy if they were given as part of CHOP according to the study drug eCRF page (EX domain).

"Study treatment" is defined as at least one dose > 0 of any component of combination therapy (e.g. obinutuzumab, atezolizumab, polatuzumab vedotin, venetoclax, lenalidomide, idasanutlin) or chemotherapy.

#### 2.2.1 Treatment Groups

The treatment arm labels to be included in the outputs are displayed as described below in following order:

Atezolizumab will be replaced by 'Atezo'

Obinutuzumab will be replaced by 'G'

Rituximab will be shown as 'R'

Polatuzumab vedotin will be replaced by 'P'

Venetoclax will be replaced by 'V'

Idasanutlin will be replaced by 'I'

Lenalidomide will be replaced by 'L'

Bendamustine will be replaced by 'B'

We also should show dose levels after each treatment. So for illustration purposes, a treatment arm of "Obinutuzumab 1000mg + Polatuzumab vedotin 1 mg/kg + Lenalidomide 10 mg" would be shown as "G (1000MG) P (1MG/KG) L (10MG)", or "Obinutuzumab 1000mg + Atezolizumab 1 mg + CHOP" would be shown as "Atezo (1MG) - G (1000MG) - CHOP".

#### 2.2.2 New Anti-lymphoma Treatment

A new anti-lymphoma treatment (NALT) is defined as any treatment reported on the 'Follow-up New Anti-Lymphoma Therapy' or 'New Anti-Lymphoma Surgery and Procedure' eCRF pages.

If a patient has more than one, use the first date from any of the NALTs.

## 2.3 Patient Allocation to Reporting Periods

The following definitions will be used to allocate AEs and laboratory data to study periods. The same definitions will also be used in other cases where applicable, e.g. patient disposition. Adverse events are assigned to the study periods based on the AE onset date.

#### 2.3.1 Study Day 1

Study day 1 is the day of first administration of any study treatment (see Section 2.2).

#### 2.3.2 Before Therapy

Any AE that occurs before study day 1 is considered to have occurred before therapy unless the end date is after the date of first study drug intake and the most extreme intensity is higher than the initial intensity (see treatment emergent rules in Section 6.2.1). For handling of pre-dose laboratory assessments, see definition of baseline (Section 2.3.3).

#### 2.3.3 Baseline

The baseline assessment is the last valid assessment in the 28 day window before first administration of a study treatment component (see Section 2.2 for study treatment definition). If no time is linked to a laboratory or vital sign assessment at study day 1, it is assumed that the assessment was done before the drug administration. For patients who never received study treatment, baseline is defined as the last valid assessment prior to or on the day of enrolment — note though that this is only applicable to parameters not being reported out using the safety population, as otherwise these patients are anyway excluded.

#### 2.3.4 Study Periods

All periods below end at the study completion or early withdrawal visit. For all periods, NALT refers to the first occurrence of NALT post study-treatment.

If a patient is ongoing in any period at the time of reporting, then consider last known alive date as the period end date just for the purpose of duration calculations and to ensure events are still mapped to this period.

#### 2.3.4.1 Treatment Period

The treatment period will be defined as the time between study day 1 and last administration of any component of the study treatment + 28 days or if a NALT starts within 28 days, then treatment period ends one day prior to the start of the NALT.

#### 2.3.4.2 Induction Treatment Period

Only relevant for studies with a maintenance or consolidation treatment period: For patients receiving maintenance or consolidation therapy, the induction treatment period will be defined as the time between study day 1 and 1 second before the first dose of maintenance or consolidation therapy, or if a NALT starts prior to the start of maintenance or consolidation, the induction treatment period ends one day prior to the start of the NALT. For those not receiving maintenance or consolidation therapy, the induction treatment period follows the same rules as given above for the treatment period (see Section 2.3.4.1).

#### 2.3.4.3 Maintenance or Consolidation Period

Only relevant for studies with a maintenance or consolidation treatment period: The maintenance or consolidation period starts on the day of the patient's first dose of any treatment in maintenance or consolidation and ends one day prior to the start of NALT or 28 days after the last dose of any maintenance or consolidation treatment.

Note: Safety outputs produced on the maintenance or consolidation period will only show the maintenance or consolidation treatment arm, and these outputs will only include those patients that enter the maintenance or consolidation period.

#### 2.3.4.4 Post treatment Follow-up Period

The follow-up period refers to the phase of the study that is post study treatment. Only patients who have an induction treatment completion eCRF page completed (for patients without a dose of maintenance or consolidation treatment) and a maintenance/consolidation treatment completion eCRF page completed (for patients who received maintenance or consolidation treatment) will be included in the follow-up period.

The follow-up period starts the day after the end of the treatment period (see Section 2.3.4.1). The follow-up period ends at the date recorded on the post treatment follow-up phase completion eCRF page, or at the last recorded date in the eCRF for patients ongoing in the period.

#### 2.3.4.5 Survival Follow-up

Survival follow-up starts the day after the follow-up period ends. Survival follow-up ends at the date recorded on the study completion/early discontinuation eCRF page, or at the last recorded date in the eCRF for patients ongoing in the period. For patients who withdrew from induction, post-induction or follow up phase due to PD, survival follow up starts the day after the date of study completion/early discontinuation.

#### 2.3.5 Treatment Cycle

A treatment cycle starts on the day of the first administration of a study treatment component and ends the second before the start of the next cycle. For example, cycle 1 will start at the first valid cycle 1 study drug administration and will end at the start date of the cycle 2 dose (or cycle 3, or 4 etc. if cycle 2 dose is missing) minus 1 second. The last cycle ends when the treatment period ends.

#### 2.3.6 Observation Time

Observation time is the time between enrolment date and the day of death or the last assessment in the database (=last known alive date, see Section 2.3.7).

#### 2.3.7 Last known alive date

The last known alive date is derived from the latest of dates in the following CRF fields: AE start and end dates (including start and end dates of IRR symptoms), tumor response assessment dates, study drug exposure dates, lab assessment dates, vital signs assessment dates, ECG assessment dates, survival follow-up pages where the status is confirmed as 'ALIVE', death date, enrolment date and date of informed consent.

As per STREAM standard rules only partial dates from tumor response or death data are included. In this case missing day is replaced by 1st of the month if only month and year are given. Dates where month and/or year are missing are not imputed but excluded. For partial death dates STREAM applies the following additional rule: If month/year of last known alive date from all other dates\* is equal to the month/year of partial death date then last known alive date is set to \* + 1 day.

#### 2.3.8 Study Drug Exposure Time

Study drug exposure time is defined as the last study treatment administration end date (where dose is > 0) minus the first study treatment administration date (where dose is > 0) plus 1 day. This could be calculated individually by study drug or collectively for all study drugs.

#### 2.3.9 General Rules

In the analysis of laboratory data by cycle, if there are several observations per cycle the last value is used. If there are two valid assessments per day and no time is available, the scheduled valid assessment will be taken. In the analysis of follow-up data by visit, patients will be assigned to visits using the clinical planned event (CPE).

All derivations of duration are initially done based on days and converted to months and years if needed using 30.4375 and 365.25, respectively, as denominator if not otherwise specified. Unless otherwise specified, months will be used in outputs.

Computation of durations: any duration in days is computed as end date minus start date + 1 day.

## 2.4 Handling of Missing and Incomplete Data

Laboratory values with either a '<' or '>' included in the lab result will have the inequality symbol removed and 0.001 will be either subtracted (when '<' is included) or added (when '>' is included) to the numeric value of the result for the purpose of summarizing (the original value will be displayed in listings). For example, laboratory values given as "<7" or ">7" are treated as follows:

| Recorded data value | When reported as numerical value | When reported in a listing |
|---|---|---|
| <7 | 6.999 | <7 |
| >7 | 7.001 | >7 |

Each AE is assigned to a time period, i.e. pre-treatment, during treatment (could be further split as induction/maintenance or consolidation) or follow-up (Section 2.3).

In listings AEs with partial dates will be shown by having a missing study day.

For AEs and concomitant treatment (not including NALTs), the following rules will be applied:

- Incomplete onset dates for AEs will be handled as follows:
  - in case the day is missing, it is replaced by the 1<sup>st</sup> of the month, unless a trial treatment exists within that month (not necessarily first treatment) then set to the date of that treatment
  - o in case the day and month are missing, they are replaced by 1<sup>st</sup> of January, unless the first trial treatment exists within that year then set to the date of that treatment
  - o in case imputation leads to the AE occurring before treatment, the onset date will be set to the treatment start date
  - resolution dates are checked to ensure imputed onset dates do not become later than the resolution date
- In case AE most extreme intensity is missing, it will be replaced by the initial intensity
- AEs with missing grades will be included in the summaries for grade 3 to 5 AEs
- AEs with missing relationship to trial medication are included in the summaries of related AEs
- AE with missing seriousness will be included in all summaries of serious adverse events (SAEs)

• For partial concomitant treatment start dates the 1<sup>st</sup> of the month will be imputed (if only day is missing) or 1<sup>st</sup> January will be imputed (if day and month are missing).

Partial dates of NALT will be imputed as follows, in order to use the most conservative (i.e. earliest) date without shortening the treatment period:

- If only the year is available then the difference between 1<sup>st</sup> January of the year and the last administration date of any component of study treatment will be checked: if the difference is >28 days then 1<sup>st</sup> January will be imputed; otherwise, if the difference is ≤28 days then the date of the last study drug administration\* + 29 days will be imputed.
- If the month and year are both available then the difference between the 1<sup>st</sup> of the month and last study drug administration will be checked: if the difference is >28 days then the 1<sup>st</sup> of the month will be imputed; otherwise, if the difference is ≤28 then the date of the last study drug administration\* +29 days will be imputed. However, if this leads to the imputed date having the month following the month in the partial date, then the last day of the partial date month will be imputed.

Partial study drug administration dates will not be imputed. A valid study drug administration record is one with a complete begin date and a >0 actual dose for antibody or chemotherapy. Only valid records should be used for all analyses where information of study drug administration is used.

Handling of partial or missing dates for other assessments are discussed within their corresponding sections.

## 3 Subgroups

Definitions of potential subgroups are included in this section. Please refer to LOPO to determine which analyses these subgroups are applied to.

#### 3.1 ABC/GCB subtypes for DLBCL patients

DLBCL cell-of-origin (COO) prognostic subgroups (ABC and GCB), defined using gene expression profiling, have been associated with different clinical outcomes in patients receiving R-CHOP for DLBCL, with GCB subgroups demonstrating a better prognosis than ABC. DLBCL patients will be classified as having the ABC or GCB cell of origin subtypes.

#### 3.2 BCL-2 subgroups for DLBCL patients

BCL-2 overexpression has been shown to have prognostic value in DLBCL DLBCL patients will be classified as having high/low BCL-2 expression.

<sup>\*</sup>For B-cell and Immunoglobulin outputs, use the last antibody administration date; for other outputs use the last of all study medication dates.

## 3.3 Double hit subgroup (FISH) for DLBCL patients

Approximately 9%–17% of patients with newly diagnosed DLBCL harbor an underlying *MYC* rearrangement, and these patients are at high risk of treatment failure with R-CHOP. A subset of patients with *MYC*-positive DLBCL also harbors an additional *BCL2* rearrangement. These "double-hit" lymphomas are associated with a very poor outcome Subgroup of 'Double hit' DLBCL patients vs. rest of DLBCL patients will be set up.

## 3.4 Double positive subgroup (IHC) for DLBCL patients

Overexpression of BCL-2 and Myc in DLBCL has also been observed in the absence of translocation. This "double-positive" DLBCL status is also associated with worse prognosis. Therefore subgroup of double positive (IHC) DLBCL patients will be set up.

Cell of Origin (COO) and BCL-2 for DLBCL patients: COO and BCL-2 based subgroups will be set up for DLBCL patients: ABC-BCL-2 high, ABC-BCL-2 low, GCB-BCL-2 high, GCB-BCL-2 low.

Cell of Origin (COO) and Myc for DLBCL patients: COO and Myc based subgroups will be set up for DLBCL patients: ABC-BCL-2 positive-MYC positive, GCB-BCL-2 positive-MYC positive.

## 3.5 IPI / FLIPI

For FL patients FLIPI based subgroups may be created. For DLBCL patients IPI based subgroups may be created.

| Applicable for Study | BO29563<br>Atezo-G-<br>B | BO29563<br>Atezo-<br>G/R-CHOP | BO29562 | BO29561 | GO29833 | GO29834 | BH29812 |
|---|---|---|---|---|---|---|---|
| ABC/GCB | | х | | х | | | Х |
| BCL-2 | | Х | | Х | | | Х |
| Double hit | | х | | х | | | х |
| Double positive | | х | | х | | | х |
| COO&Myc | | х | | х | | | Х |
| MRD | Х | х | Х | х | | | Х |
| IPI/FLIPI | х | х | х | х | | | х |
| p53 | | | | | | | х |
| CD8 | х | Х | Х | х | | | |
| PDL1 | х | х | х | х | | | |
| CD58 | | х | | | | | |
| CD79 | | | | х | | | |

# 4 Demographics, Baseline Disease Characteristics and Prognostic Markers

## 4.1 Demographics

Demographics are collected at enrollment and generally may include:

- Gender
- Age at BL
- Race
- Ethnicity
- Weight
- Height
- BMI (= body mass index)
- BSA (= body surface area)
- ECOG Performance score at BL

## 4.2 Baseline Disease Characteristics and Prognostic Markers

Baseline Disease Characteristics and Prognostic Markers are baseline conditions specifically related to the indication under study. These may include:

- Histology/pathologic diagnosis
- Ann Arbor stage
- Time since first histologic or pathologic diagnosis
- Biomarker status from tumor tissue or blood samples at BL
  - o COO
  - o BCL-2
  - o MYC
  - o COO and BCL-2
  - o BCL-2 and MYC(FISH)
  - o BCL-2 and MYC(IHC)
  - o COO and BCL-2 and MYC

- o P53 (in studies with idasanutlin)
- IPI
- FLIPI
- Follicular Lymphoma Grade
- Any B symptoms at BL
- Individual B-symptoms, i.e. fever, weight loss, night sweats, at BL
- Bulky disease (threshold 70 mm) at BL
- Number of Indicator Lesions at BL
- Number of non-Indicator Lesions at BL
- Spleen Assessment at BL: Palpable yes/no or >13 cm in vertical length vs. <=13 cm (r/r DLBCL/FL)</li>
- Liver Assessment at BL: Palpable yes/no
- SPD of Indicator Lesions at BL
- Number of prior anti-lymphoma therapies
- Prior radiotherapies
- Prior surgeries or procedures
- Serum LDH at BL(>normal vs. <=normal)</li>
- Extranodal Involvement at BL yes/no
- If yes, Number of extranodal sites at BL
- Bone Marrow Involvement
- Status (relapsed/refractory or previously untreated) (BO29563)
- PET score at BL
- Presence of FDG avid lesions representing lymphoma at BL yes/no (detected by PET scan)
- Evidence of FDG avid disease in bone marrow at BLyes/no (detected by PET scan)

## **5 Efficacy Analyses**

The efficacy analyses will be performed on the efficacy evaluable population, which includes all patients who received at least one dose of any components of the combination during the expansion

phase. Patients who received any study drugs at the RP2D during the dose-escalation/safety run-in phase may be pooled with the efficacy evaluable population depending on protocol.

For studies which have specific definition of the efficacy population, refer to protocol for the definition. For example, Study BH29812: The primary and secondary efficacy analyses will include all patients enrolled in the expansion phase.

## 5.1 Analysis of Primary Endpoint

The primary efficacy endpoint is the proportion of patients achieving a CR at EOI, as determined by the IRC on the basis of PET-CT scans according to modified Lugano 2014 criteria. Point estimates will be presented, along with the corresponding 90% Clopper-Pearson exact CIs. Patients without a post-baseline tumor assessment will be considered non-responders.

## 5.2 Analysis of Secondary Endpoints

The secondary efficacy analyses will be estimation of the proportion of patients who achieve each of the following endpoints:

- CR at EOI, as determined by the investigator on the basis of PET-CT scans
- CR at EOI, as determined by the IRC and by the investigator on the basis of CT scans alone
- Objective response (defined as a CR or PR) at EOI, as determined by the IRC and by the investigator on the basis of PET-CT scans
- Objective response (defined as a CR or PR) at EOI, as determined by the IRC and by the investigator on the basis of CT scans alone
- Best response of CR or PR during the study, as determined by the investigator on the basis of CT scans alone

#### Study BO29563:

- CR at EOI, as determined by the investigator on the basis of PET-CT scans using modified Lugano 2014 criteria
- CR at EOI, as determined by the IRC and by the investigator on the basis of PET-CT and CT scans using modified Cheson 2007 criteria
- Objective response (defined as a CR or PR) at EOI, as determined by the IRC and by the investigator using modified Lugano 2014 criteria and modified Cheson 2007 criteria
- Best objective response (defined as a CR or PR) during the study (including all tumor assessments), as determined by the investigator using modified Cheson 2007

Point estimates will be presented, along with the corresponding two-sided 90% Clopper-Pearson exact CIs. Patients without a post-baseline tumor assessment will be considered non-CRs and non-responders, respectively.

## 5.3 Analysis of Exploratory Endpoints

Exploratory efficacy analyses will include estimation of the proportion of patients achieving each of the following endpoints:

- For patients who have positive PET scans at EOI: CR at 12 months, as determined by the IRC and by the investigator on the basis of PET-CT scans
- CR at 12 months, as determined by the investigator on the basis of CT scans alone (BO29561)
- CR at 12, 24, and 30 months in patients with previously untreated FL, as determined by the investigator using modified Cheson 2007 criteria (BO29563)
- Additional descriptive analysis based on TP53 status will be performed on the following endpoint: CR at EOI, as determined by the IRC on the basis of PET-CT scans (BH29812)

Point estimates will be presented, along with the corresponding two-sided 90% Clopper-Pearson exact CIs. Patients without a post-baseline tumor assessment will be considered non-CRs and non-responders, respectively.

Exploratory efficacy analyses will also be performed on the following endpoints:

- PFS, defined as the time from initiation of study treatment to first occurrence of disease progression or relapse, as determined by investigator on the basis of CT scans alone, or death from any cause
- EFS, defined as the time from initiation of study treatment to any treatment failure, including disease progression or relapse, as determined by investigator on the basis of CT scans alone, initiation of new anti-lymphoma therapy, or death from any cause, whichever occurs first
- DFS, defined, among patients achieving a CR, as the time from the first occurrence of a
  documented CR to relapse, as determined by the investigator on the basis of CT scans alone, or
  death from any cause, whichever occurs first
- DOR, defined as the time from the initial response to disease progression or death among patients who have experienced a CR or PR during study (Study BO29561/BO29562).
- OS, defined as the time from initiation of study treatment to death from any cause

PFS, EFS, DFS, DOR, and OS will be summarized descriptively using the Kaplan-Meier method (Kaplan and Meier 1958). For the PFS, EFS, and DFS analyses, data for patients without an event of interest will be censored at the date of the last tumor assessment. For the PFS and EFS analyses, data for patients without post-baseline tumor assessments will be censored at the date of initiation of study treatment plus 1. For the DFS analysis, data for patients without a tumor assessment after the first CR will be censored at the date of first CR tumor assessment + 1 day. For the DOR analysis, data for patients without a tumor assessment after the Objective Response (OR) of CR or PR will be censored at the date of OR tumor assessment +1 day. For the OS analysis, data for patients who have not died will be censored at the date the patient was last known to be alive. Where medians are reached, the corresponding estimated median will be provided, along with the 95% CI using the method of

Brookmeyer and Crowley (1982). In addition, landmark estimates of the proportion of patients who are event free at 6 months, 9 months, 1 year, and 2 years will be provided, along with 95% asymptotic CIs using Greenwood's formula for standard errors.

#### 5.4 Interim Analyses

It is anticipated that at least one interim analysis will be conducted during the expansion phase of the study, when at least 15 patients in one treatment arm have been evaluated for PET-CT—defined CR at the EOI.

## 6 Safety Analyses

Safety analyses will be based on all patients who received at least 1 component of study medication. For safety analyses, patients will be reported by the treatment actually received. Patients who only received certain treatments from a combination group, but not all, will be reported by the planned treatment group.

Study data will be summarized separately for each phase. Data from the dose-escalation/safety runin phase will be summarized by cohort (assigned dose level). Data from the expansion phase will be summarized by histological subtype (i.e., FL or DLBCL) and treatment group if applicable.

#### 6.1 Exposure

Exposure summaries will be done by study period, i.e. there will be separate outputs for induction and post-induction phase. Exposure summaries will also be done by cycle if necessary.

#### 6.1.1 Extent of Exposure to Study Drug

At least one component of study treatment (i.e. obinutuzumab, rituximab, atezolizumab, polatuzumab vedotin, venetoclax, lenalidomide, idasanutlin or chemotherapy as defined in section 2.2) per cycle requires a received dose of >0 to be considered as a received cycle.

#### 6.1.2 Dose Intensity

The dose intensity will be calculated based on the total received dose as compared to total planned dose (based on planned dose of first intake). Patients who withdrew prematurely from one study drug component but are still receiving other components of the study drug will be included in the calculation of the dose intensity up until the last day on which they received any study drug component.

E.g a patient in Atezo-G-Benda arm in BO29563 in induction had 5 doses of G with last dose on Cycle 3 Day 1, and 7 doses of Bendamustine with last dose on Cycle 4 Day 1. Number of expected doses for G would be 6, dose intensity for G would be 5 \* 1000 mg / 6 \* 1000 mg.

The intensity categories are: <60%, 60 - <80%, 80 - <90%, >=90%, Missing. Summary statistics (mean, s.d., median, range) will also be used to summarize the dose intensity.

Dose intensity will be summarized separately for the induction and post-induction phase. For drugs in Prednisone category in BO29563, i.e. Methylprednisolone, Prednisone, Prednisolone and Dexamethasone, dose intensity is calculated for the whole category as number of actually received doses divided by number of expected doses up to the last time point any component of study drug was received.

#### 6.2 Adverse Events

#### 6.2.1 General AE Reporting

Listings will include all AEs. A flag will indicate to which study period an AE is assigned to: before treatment, initial/induction treatment, maintenance/consolidation treatment or follow up.

Study periods are as defined in Section 2.3.4. An AE is assigned to a period using the AE onset date, Unless otherwise specified, AE and SAE summary tables will be restricted to those that are treatment emergent, defined as starting on or after the day of first dose of any drug. For summary tables on the follow-up period, no upper time window is implemented, that is, all AEs from start of follow-up onwards will be included.

Generally AE will be summarized by study period.

In addition selected adverse events and AESI (see categories in subsequent tables) may be summarized by treatment cycle. An AE will be assigned to a cycle based on the AE onset day relative to cycle start day. Cycle start day is the first day on which any study medication was administered. AEs with onset on cycle start day will be included in the respective cycle.

In studies BO29561, BO29562 and BO29563 AESI based on tickbox in CRF page and on causality to any study drug will be reported separately .

#### 6.2.2 Selected AEs and AE of Special Interest (AESI)

Selected AE and AESI were defined based on the clinical experience with study treatment components that represent an IMP. Also anticipated potentially overlapping toxicities as specified in respective study protocols need to be taken into account.

Definitions for selected AE and AESI are provided in subsequent tables.

| Selected AE Category | Definition | BO29563 | BO29562 | BO29561 | BH29812 | BH39147 | GO29833 | GO29834 |
|---|---|---|---|---|---|---|---|---|
| Thrombocytopenia | SMQ "HAEMATOPOIETIC<br>THROMBOCYTOPENIA narrow"<br>(20000031n) | х | х | х | х | х | х | х |
| Hepatitis B reactivation/newly occurring | PT 'HEPATITISB' | х | х | x | х | х | х | х |
| Cardiac AE | SOC "CARDIAC DISORDERS" | х | х | х | x | х | х | х |
| Infusion Related Reaction (IRR) | PT 'INFUSION RELATED REACTION' and related to at least one component of study treatment and event occurred within 24 hours or during infusion and tickbox 'Systemic Infusion Reaction' ticked (This definition was applied in BO29563- study lead BioStats/SPA please check if this is valid for your study) | x | x | x | x | x | x | x |
| Infections | SOC 'INFECTIONS AND INFESTATIONS' | х | х | х | х | X | х | х |
| Neutropenia | Roche Standard AEGT "NEUTROPENIA AND ASSOCIATED COMPLICATIONS" (for BO29561- 3:including late onset and prolonged neutropenia) (SMQ Haematopoietic leukopenia narrow for GO29833/834) | х | х | х | х | х | х | х |

| Selected AE Category | Definition | BO29563 | BO29562 | BO29561 | BH29812 | BH39147 | GO29833 | GO29834 |
|---|---|---|---|---|---|---|---|---|
| Prolonged neutropenia | Initial ANC < 1.0 × 109/L that is<br>still present 28 days after<br>treatment with GA101 | | | | х | x | | |
| Late onset Neutropenia | ANC < 1.0 × 109/L occurring >= 28<br>days after ga101 infusion has been<br>completed/stopped | | | | х | X | | |
| Gastrointestinal perforation | SMQ "GASTROINTESTINAL<br>PERFORATION" (20000107<br>narrow). | x | х | х | x | x | х | x |
| Peripheral Neuropathy<br>(motor/and or sensory) | SMQ Peripheral neuropathy<br>wide | | | x | | | х | х |
| Dose Limiting Toxicity | CRFtickbox | | | | х | | | |
| Drug-drug interactions | Single PT | | х | | | | | |

| AE of Special Interest | Definition | BO29563 | BO29562 | BO29561 | BH29812 | BH39147 | GO29833 | GO29834 |
|---|---|---|---|---|---|---|---|---|
| Drug induced liver injury | Respective tickbox for AESI on<br>CRF page ticked | | | | x | x | х | х |
| Suspected transmission of infectious agent | Respective tickbox for AESI on<br>CRF page ticked | | | | х | х | х | х |
| Grade 4 thrombocytopenia | SMQ "HAEMATOPOIETIC<br>THROMBOCYTOPENIA narrow"<br>(20000031n) | | | | | | x | |
| Grade≥ 3 infection | SOC | | | | | | x | |
| Grade ≥ 3 thrombocytopenia<br>or Grade 2 thrombocytopenia<br>if associated with<br>hemorrhage/bleeding | ? | | | | х | x | | |
| Grade ≥ 2 diarrhea | ? | | | | X | Х | | |
| Grade≥3 neutropenia,<br>including febrile neutropenia | SMQ HAEMATOPOIETIC<br>LEUKOPENIA (narrow) | | | | х | x | | |
| Grade ≥ 2 C. difficile infection | ? | 9 | 9 | | X | х | | |
| Immune-related Pneumonitis | SMQ INTERSTITIAL LUNG DISEASE (narrow) | х | X | х | | | | |
| Immune-related Colitis | HLT COLITIS (excluding infective) | х | х | х | | | | |
| Immune-related Adrenal insufficiency | AEGT Atezolizumab<br>comprehensive adrenal<br>insufficiency search - 22 Jul<br>2015 | х | х | х | | | | |
| Immune-related Diabetes<br>Mellitus | AEGT Atezolizumab<br>Diabetes/DKA (excludes<br>Hyperglycemia) | Х | X | Х | | | | |

| AE of Special Interest | Definition | BO29563 | BO29562 | BO29561 | BH29812 | BH39147 | GO29833 | GO29834 |
|---|---|---|---|---|---|---|---|---|
| Immune-related Pancreatitis | ATEZOLIZUMAB PANCREATITIS<br>AEGT | х | х | х | | | | |
| Immune-related hypothyroidism | Hypothyroidism SMQ (wide) | х | x | х | | | | |
| Immune-related<br>hyperthyroidism | Hyperthyroidism SMQ (narrow) | х | x | х | | | | |
| Immune-related Hepatitis | HEPATIC FAILURE, FIBROSIS AND CIRRHOSIS AND OTHER LIVER DAMAGE-RELATED CONDITIONS SMQ (narrow); HEPATITIS NON-INFECTIOUS SMQ (narrow); LIVER RELATED INVESTIGATIONS, SIGNS AND SYMPTOMS SMQ (narrow) | x | x | x | | | | |
| Immune-related Guillain-Barré<br>syndrome | GUILLAIN-BARRE SMQ (narrow) | х | X | X | | | | |
| Immune-related Myasthenia gravis | HLT MYASTHENIA GRAVIS AND RELATED CONDITIONS | х | х | х | | | | |
| Immune-Related Nephritis | HLT glomerulonephritis and<br>nephrotic syndrome or HLT<br>nephritis NEC | х | х | х | | | | |
| Immune-related Meningitis | Noninfectious meningitis SMQ (narrow | х | x | х | | | | |
| Immune related Encephalitis | Noninfectious encephalitis<br>SMQ (narrow) | x | x | x | | | , | |
| Immune-related myositis | HLT muscle infections and inflammations; HLT muscular autoimmune disorders | х | х | х | | | | |

| AE of Special Interest | Definition | BO29563 | BO29562 | BO29561 | BH29812 | BH39147 | GO29833 | GO29834 |
|---|---|---|---|---|---|---|---|---|
| Immune-related<br>Rhabdomyolysis | SMQ Rhabdomyolysis /<br>myopathy (narrow) | х | х | х | | | | |
| Immune-related Rash | AEGT EGFR Associated Skin<br>Reactions | x | x | х | | | | |
| IRR/Hypersensitivity Infusion<br>Related Reactions | AEGT Kadcyla specific AEGT Infusion Related reactions/Hypersensitivity (type 1) 14 Feb 2013 PTs 'Infusion Related Reaction', 'Cytokine Release Syndrome' Only AE with onset on same day or within 1 day of Atezo infusion are flagged | x | x | x | | | | |
| Systemic immune Activation | Systemic Immune Activation<br>(PT), Cytokine Release<br>Syndrome (PT) | X | х | х | | | , | |
| Immune Related Ocular Inflammatory Toxicity | AEGT ATEZOLIZUMAB OCULAR INFLAMMATION TOXICITY) | Х | Х | X | | | | |
| Immune-related Vasculitis | Vasculitis (SMQ) narrow | х | X | х | | | | |
| Immune-related Hypophysitis | hypothalamic and pituitary<br>disorders NEC (HLT) | х | х | х | | | | |
| Immune-related Myocarditis | Noninfectious myocarditis<br>(HLT), Noninfectious<br>pericarditis(HLT), Cardiac<br>failure (SMQ) narrow AEGT<br>Atezolizumab Myocarditis<br>Immune Related | х | х | х | | | | |

| AE of Special Interest | Definition | BO29563 | BO29562 | BO29561 | BH29812 | BH39147 | GO29833 | GO29834 |
|---|---|---|---|---|---|---|---|---|
| Immune-related Severe Cutaneous Reaction | Severe cutaneous adverse reactions (SMQ) narrow | x | х | х | | | | |
| Secondary malignancy | "Malignant or Unspecified<br>Tumours" (2000009w), starting<br>6 months after the first study<br>drug intake or later | х | х | х | х | х | х | х |
| Tumor Lysis Syndrome | PT: 'TUMOUR LYSIS<br>SYNDROME' | х | х | х | х | х | х | х |
| Auto-Immune Hemolytic<br>Anaemia | Haemolytic Disorders (SMQ) narrow | x | x | х | | | | |

PT = Preferred Term, HLT = High Level Term, HLGT = High Level Group Term, SOC = System Organ class, SMQ=Standard MedDRA Queries

For Atezo specific AESI (i.e. all categories of AESI listed in table except secondary malignancy and TLS) only AE with causality to Atezo suspected and onset on or after start of cycle 2 are considered.

#### 6.3 Concomitant Medications

Outputs for concomitant medications will include any treatment reported on the "Concomitant Medications" form eCRF pages, with additional pages included as required per study. Prophylactic medication and premedication, such as anti-coagulant agents including aspirin and LMWHs, will be summarized separately.

#### 6.3.1 Corticosteroids

For any analyses requiring identification of corticosteroids we will use the company standard 'corticosteroids' drug basket created by the Drug Basket Committee (DBC) at: <a href="http://we2.collaboration.roche.com/team/2012137a/SitePages/Default.aspx">http://we2.collaboration.roche.com/team/2012137a/SitePages/Default.aspx</a>. We will use the full list of terms from this basket.

For atezolizumab contained studies, impact of steroids on atezolizumab and IRR prevention will be explored.

#### 6.4 Laboratory Data

Laboratory data that have been obtained will be converted to System International (SI) units. Grading system will be from NCI-CTC version 4. Where normal ranges are required to be converted, the Roche References Ranges will be used (cf. gcp spt000144). The grading will be defined as follows:

#### Project-specific Gradings:

| Parameter | SI Unit | Grade 4 Low | Grade 3 Low | Grade 2 Low | Grade 1 Low |
|---|---|---|---|---|---|
| LYMPH | 10**9/L | < 0.2 | 0.2 to < 0.5 | 0.5 to < 0.8 | 0.8 to < 1 |
| NEUTR | 10**9/L | < 0.5 | 0.5 to < 1 | 1 to < 1.5 | 1.5 to < 1.8 |
| CRCL | mL/min | < 15 | 15 to < 30 | 30 to < 60 | 60 to < LLN |

| Parameter | SI Unit | Grade 1 High | Grade 2 High | Grade 3 High | Grade 4 High |
|---|---|---|---|---|---|
| LYMPH | 10**9/L | - | > 4 to 20 | > 20 | - |
| NEUTR | 10**9/L | - | - | - | - |
| CRCL | mL/min | - | - | - | - |

#### 6.4.1 Hematology and Chemistry Laboratory Data

Summary tables will be produced for the hematology and chemistry laboratory parameters (LBCAT=HEMATOLOGY, LBCAT=CHEMISTRY).

#### 6.4.2 General Derivation Rules on Absolute Counts/Percentages

The laboratory parameters such as lymphocytes, eosinophils, basophils and monocytes might be recorded as absolute count or percentage in the eCRF. If on the same day and time, the absolute count

of the laboratory parameter is missing but the percentage is not missing, then the absolute count will be derived from the percentage to absolute count as follows:

ABSOLUTE\_COUNT = PERCENTAGE x WBC, where WBC is white blood cell (LBTESTCD=WBC) and expressed as cells per microliter (LBSTRESU =  $10^9$ /L, or  $10^3$ /uL). Note that WBC values collected on the same date and time will be used in the derivation of absolute count. If the WBC value is missing on the same day and time then the absolute count of the laboratory parameter will also be missing.

Note: If a patient has multiple values of the same assessment on the same day and at the same time, the minimum values recorded will be retained for the calculation of the absolute counts.

#### 6.4.3 Absolute Neutrophil Counts

Neutrophil count recovery is defined as absolute neutrophil count ANC  $\geq 1.0 \times 10^9$ /L, given ANC was collected after the patient has had his last dose of antibody, and ANC <  $1.0 \times 10^9$ /L at the last previous visit before EOT. Neutrophil count recovery (ANC  $\geq 1.0 \times 10^9$ /L) should not be immediately followed by ANC <  $1.0 \times 10^9$ /L, or a missing assessment, but only by ANC  $\geq 1.0 \times 10^9$ /L at the next visit.

| VISIT 1 | VISIT 2 | VISIT 3 | VISIT 4 | OUTCOME |
|---|---|---|---|---|
| $< 1.0 \times 10^{9}/L$ | $\geq$ 1.0 $\times$ 10 $^{9}$ /L | missing | missing | Not |
| | | | | RECOVERED |
| < 1.0 × 10 <sup>9</sup> /L | $\geq$ 1.0 $\times$ 10 $^{9}$ /L | $\geq$ 1.0 $\times$ 10 $^{9}$ /L | $< 1.0 \times 10^{9}/L$ | RECOVERED |
| < 1.0 × 10 <sup>9</sup> /L | $\geq$ 1.0 $\times$ 10 $^{9}$ /L | < 1.0 × 10 <sup>9</sup> /L | < 1.0 × 10 <sup>9</sup> /L | NOT |
| | | | | RECOVERED |
| < 1.0 × 10 <sup>9</sup> /L | $\geq$ 1.0 $\times$ 10 $^{9}$ /L | missing | < 1.0 × 10 <sup>9</sup> /L | NOT |
| | | | | RECOVERED |

Time to neutrophil count recovery is defined as the number of days between the date of last dose of antibody and the date of single recovery. In case a patient was not depleted at last dose of antibody, no time to single recovery will be calculated. Where no ANC value occurs at the last drug intake, the next valid ANC assessment will be taken. For instance, ANC values at the EOT visit might be used instead if there is no ANC assessment on the day of the last dose of the antibody. If there are multiple ANC records at a visit, the last ANC assessment will be retained provided there is a valid identifier. If a study does not have a valid identifier, the lowest ANC value at the visit will be used instead.

#### 6.4.4 Serum Creatinine Clearance

Serum creatinine clearance will be derived using the Cockcroft-Gault formula (where needed).

#### 6.4.5 Hy's Law Cases

Patients with ALT > 3x BL OR AST > 3x BL AND Total Bilirubin >2xULN within 14 days, at any time for post baseline measurement, will be investigated for potential Hy's Law cases in a patient listing.

A summary table showing the proportion of patients with elevated ALT, AST, ALP and Total Bilirubin will also be produced.

#### 6.4.6 B-Cell Depletion and Recovery

B-cell depletion is defined as CD19 B-cell count  $< 0.07 \times 10^9 / L$  and can only occur after at least one dose of antibody has been administered.

Time to depletion is defined as the number of days between the first intake of study drug and the date of first depletion (assessments at study day 1 after start of the infusion are considered as after baseline).

Note that CD19 B-cells with no time record are assumed to be collected before the first treatment dose. Hence B-cells with no associated time that are collected on the same day as the last dose of the antibody will be assumed to be pre-dose.

#### 6.4.6.1 B-cell recovery

B-cell recovery is defined as CD19 B-cell count >= 0.07x109/L, and B-cell was collected after LAA, the patient's B-cells were previously depleted and recovery is not followed exclusively by further depletion, i.e. B-cell recovery at a visit cannot be immediately followed by B-cell depletion, or a missing assessment, but only by recovery at the next visit. Assuming the situation 4 B-cell assessments at 4 visits:

| VISIT 1 | VISIT 2 | VISIT 3 | VISIT 4 | OUTCOME |
|----------|-----------|-----------|----------|-----------|
| DEPLETED | RECOVERED | missing | missing | Not |
| | | | | RECOVERED |
| DEPLETED | RECOVERED | RECOVERED | DEPLETED | RECOVERED |
| DEPLETED | RECOVERED | DEPLETED | DEPLETED | NOT |
| | | | | RECOVERED |
| DEPLETED | RECOVERED | missing | DEPLETED | NOT |
| | | | | RECOVERED |

Time to B-cell recovery is defined as the number of days between the date of LAA and the date of single recovery. In case a patient was not depleted at last dose of antibody, no time to single recovery will be calculated. Where no CD19 value occurs at LAA, the next valid CD19 assessment will be taken. For instance, CD19 values at the EOT visit might be used instead if there is no CD19 assessment on the day of LAA. If there are multiple CD19 records at a visit, the last CD19 assessment will be retained provided there is a valid identifier. If a study does not have a valid identifier, the lowest CD19 value at the visit will be used instead.

The Nadir is the lowest absolute CD19 value for the patient across all visits after baseline (assessment at study day 1 after start of the infusion is considered as after baseline). The time to nadir is the study

day of the earliest occurrence of the nadir value. In case of consecutive visits with the same value, the earliest date of assessments will be used. The time to nadir will be calculated as the study day of the earliest occurrence of the nadir value.

The parameters to be summarized will be CD19 + B-cell depletion and recovery over time, time to depletion, duration of depletion, time to recovery, and time to follow up without recovery.

Disease progression will be taken into account in the summary of B-cell recovery: patients with PD before B-cell recovery or PD within 45 days after recovery will be accounted for in 'Recovery with PD'; other patients will accounted for in 'Recovery without PD'. Time to B-cell recovery will be summarized separately for all patients and for patients who were in response at the time of recovery (no PD before or within 45 days from recovery). Patients with PD before recovery or within 45 days after recovery will be censored at the minimum of progressive disease date and B-cell recovery date.

B-cell depletion and recovery will be assessed up to the first day of NALT. Missing CD19 values might be recorded as "NOT DONE" or ".".

#### 6.4.7 T cell and NK cell counts

The summary of the mean (+/-SD) for the T cell (CD3, CD4, CD8) and NK cell counts (CD16 and CD56) will be shown over time in a figure where T-cell and NK-cell data are available.

#### 6.4.8 PD-L1 (CD274), PD-1, B7-1 (CD80)

The appropriate outputs, summary or listing, will be produced for studies with atezolizumab.

#### 6.4.9 Pharmacokinetik Samples, HAHA, HACAand ATA

PK serum concentration of obinutuzumab, atezolizumab, lenalidomide, polatuzumab vedotin, venetoclax, Idasanutlin will be analysed. Immunogenicity to obinutuzumab, atezolizumab, Rituximab and polatuzumab vedotin will be explored analytically based on the immune response relative to the HAHA, HACA or ATA prevalence at baseline.

#### 6.4.10 Immunoglobulins

#### 6.4.10.1 Immunoglobulin Depletion and Recovery

Immunoglobulin depletion and recovery during follow up will be derived according to the following:

## Lower immunoglobulin thresholds:

o IgA: 0.5 g/L

IgM: 0.3 g/L

o IgG: 5 g/L

#### Depletion after Baseline:

- YES = (Lab value < Lower Threshold)</li>
- NO = (Lab value >= Lower Threshold)

#### Recovery:

- YES = (Lab value >= Lower Threshold), and the lab value was collected after the last dose of antibody and patient was previously depleted
- NO = (Lab value < Lower Threshold) and the lab value was collected after the last dose of antibody and patient was previously depleted (only displayed for last value in patient listing)

Recovery (single) is the first recovery based on definition above which is not followed exclusively by further depletion i.e. recovery at a visit cannot be immediately followed by depletion, or a missing assessment, but only by recovery at the next visit. Time to single recovery is defined as the number of days between the date of last dose of antibody and date of single recovery. In case a patient was not depleted at the last dose of antibody no time to single recovery will be calculated. Where no immunoglobulin value occurs at the last dose of antibody, the next valid immunoglobulin assessment will be taken. If there are multiple immunoglobulin records at a visit, the last immunoglobulin assessment will be retained provided there is a valid identifier. If a study does not have a valid identifier, the lowest immunoglobulin value at the visit will be used instead. Recovery will be assessed up to the first day of NALT.

Analysis will be done separately for IgA, IgM and IgG. No time windows will be applied. Only visits with a valid date and non-missing values will be considered for the derivation of immunoglobulin recovery and depletion. Immunoglobulins with no associated time that are collected on the same day as the last dose of the antibody will be assumed to be pre-dose.

Descriptive statistics (n, mean, sd, median, range) will be produced at each timepoint where immunoglobulin values are available to describe the course of IgA, IgG and IgM.

An output will be produced to look at the proportion of patients with low immunoglobulin levels at each timepoint where immunoglobulin values are available.

# 7 Pharmacokinetic Analyses

PK analyses will be defined in a separate analysis plan.

## **8 Protocol Deviations**

Major protocol deviations will be taken from the PDMS system. All major deviations from PDMS will be listed and summarized and will be reported in the CSR.

## 9 References

# 10 Output Template

This section will contain all output templates, including those produced by STREAM.

# 10.1 Output 1 Enrollment by Country and Investigator

| Country,<br>Investigator Number / Name | Treatment<br>Group 1 (N=nn) | Treatment<br>Group 2 (N=nn) |
|---|---|---|
| - 01 0 | | v 200 |
| Country 1 | nn (xx.x%) | nn (xx.x%) |
| xxxxx / LastName, FirstName | nn (xx.x%) | nn (xx.x%) |
| xxxxx / LastName, FirstName | nn (xx.x%) | nn (xx.x%) |
| *** | | |
| Country 2 | nn (xx.x%) | nn (xx.x%) |
| xxxxx / LastName, FirstName | nn (xx.x%) | nn (xx.x%) |
| *** | | |

## Programming notes:

1. Analysis population: ITT

2. Template ID: ENT02

3. Program name: T\_EN

## 10.2 Output 2 Patient Disposition

| Status | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Alive on Induction Phase | nn (xx.x%) | nn (xx.x%) |
| Alive on Maintenance/Consolidation<br>Phase | nn (xx.x%) | nn (xx.x%) |
| Alive in follow-up | nn (xx.x%) | nn (xx.x%) |
| Discontinued study | nn (xx.x%) | nn (xx.x%) |
| Reason 1 | nn (xx.x%) | nn (xx.x%) |
| Reason 2 | nn (xx.x%) | nn (xx.x%) |
| Reason 3 | nn (xx.x%) | nn (xx.x%) |
| Reason 4 | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |

#### Programming notes:

- 1. Analysis population: ITT
- 2. Template ID: DST01
- 3. Program name: T\_DS
- 4. CRF: Study Drug Administration, Maintenance Phase Completion, Consolidation Phase Completion, Study Drug Discontinuation
- Alive on induction phase: subject took at least one dose of study medicine and
  was on induction phase (at least one study treatment Induction Phase
  Completion or discontinuation was **not** recorded AND study treatment
  discontinuation was **not** recorded on eCRF)
- 6. Alive on maintenance/consolidation phase: subject took at least one dose of study medicine on maintenance/consolidation phase and was on maintenance/consolidation phase (at least one maintenance study treatment discontinuation was **not** recorded and study discontinuation was **not** recorded on eCRF)
- 7. Alive in follow-up: all study treatment discontinuation was recorded but study discontinuation was **not** recorded on eCRF
- 8. Discontinued study: study discontinuation was recorded on eCRF
- 9. For BH29812, no maintenance/consolidation for DLBCL patients

# 10.3 Output 3 Analysis Populations

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| ITT (Enrolled Population) | | |
| Safety Evaluable Population | | |
| Total Exclusions | | |
| Reason 1 | | |
| Reason 2 | | |
| Efficacy Evaluable Deputation | | |
| Efficacy Evaluable Population | | |
| Total Exclusions | | |
| Reason 1 | | |
| Reason 2 | | |

# 10.4 Output 4 Listing of Patients Excluded from Analysis Populations



# 10.5 Output 5 Study Drug Completion Status and Reasons of Withdrawals from Study Drug

| Status | Treatment | Treatment Group |
|---|---|---|
| Status | Group 1 (N=nn) | 2 (N=nn) |
| Induction Phase | | at an analysis of Paragraphy & Maria |
| Discontinued study drug 1 | nn (xx.x%) | nn (xx.x%) |
| Reason 1 | nn (xx.x%) | nn (xx.x%) |
| Reason 2 | nn (xx.x%) | nn (xx.x%) |
| Reason 3 | nn (xx.x%) | nn (xx.x%) |
| Reason 4 | nn (xx.x%) | nn (xx.x%) |
| 255 | nn (xx.x%) | nn (xx.x%) |
| Discontinued study drug 2 | nn (xx.x%) | nn (xx.x%) |
| Reason 1 | nn (xx.x%) | nn (xx.x%) |
| Reason 2 | nn (xx.x%) | nn (xx.x%) |
| *** | nn (xx.x%) | nn (xx.x%) |
| Maintenance/Consolidation Phase | | |
| Discontinued study drug 1 | nn (xx.x%) | nn (xx.x%) |
| Reason 1 | nn (xx.x%) | nn (xx.x%) |
| Reason 2 | nn (xx.x%) | nn (xx.x%) |
| ••• | nn (xx.x%) | nn (xx.x%) |

## Programming notes:

1. Analysis population: Safety

2. Template ID: DST01

3. Program name: T\_DS\_DRG

1. CRF: Study Drug Administration

## 10.6 Output 6 Duration on Treatment and Follow-up

| | Treatment Group<br>1 (N=nn) | Treatment Group<br>2 (N=nn) |
|---|---|---|
| Duration on Treatment (months) | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x |
| Min-max | xx–xx | xx-xx |
| Duration of Study Period (months) | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-max | xx-xx | xx-xx |

Duration on Treatment was calculated as time from the first dose date until the last dose date + 1 day. Patients without any study medication were excluded.

Duration of Study Period was calculated as time from the first dose date to the last dates the patients were known to be alive or their death dates if died + 1 day.

Programing notes:

1. Analysis population: Safety

2. Template ID: DMT01

3. Program name: T DS DUR

4. Use descriptive method

5. CRF: Study Drug Administration

6. Duration of study period: Patients for whom no death is captured on the clinical database use the date they were known to be alive (see Section 2.3.7).
Output 7 Listing of Patients Who Discontinued Early from Study Drug

| Center/<br>Patient ID | Age/Sex/Race | Drug* | Date of First<br>Study Drug<br>Administration | Day of Last<br>Study Drug<br>Administration | Day of Study<br>Discontinuation* | Reason for<br>Discontinuation<br>from study drug* | Reason for<br>Discontinuation<br>from study |
|---|---|---|---|---|---|---|---|
| | | Treatment1 | | 12 | 14 | Adverse event | Adverse event |
| | | Treatment2 | | 36 | 65 | Lost to follow-up | Lost to follow-up |
| | | Treatment3 | | 36 | 65 | Lost to follow-up | Lost to follow-up |

#### Programing notes:

1. Analysis population: Safety

2. Template ID: DSL02

3. Program name: L\_DS\_DRG

4. Reason for Discontinuation from study: leave blank if a patient discontinued from study drug but not discontinued from study

5. Date of first study drug administration: use the first date of any drug

6. Day of last study drug administration: use the day for the certain drug

7. \*: one line for each drug

# 10.8 Output 8 Major Protocol Deviations

| | Treatment Group<br>1 (N=nn) | Treatment Group 2 (N=nn) | | | |
|---|---|---|---|---|---|
| Total number of patients with at least one major | nn (xx.x%) | nn (xx.x%) | | | |
| Proto col Deviation | | | | | |
| Total number of major protocol deviations | nn | nn | | | |
| Inclusion Criteria | | | | | |
| Age criteria | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Exclusion Criteria | | | | | |
| Pregnancy criteria | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Sodium > 180mg | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Procedural | | | | | |
| Incorrect dose | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

### Programing notes:

1. Analysis population: ITT

2. Template ID: PDT01

3. Program name: T\_DV

# 10.9 Output 9 Listing of Major Protocol Deviations



- 1. Analysis population: ITT
- 2. Program name: L\_DV

10.10 Output 10 Demographics and Baseline Characteristics

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Age (yr) | 100 | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x |
| Min-max | xx-xx | xx-xx |
| Age group (yr) | | |
| n | nnn | nnn |
| 18 <del>-4</del> 0 | nn (xx.x%) | nn (xx.x%) |
| 41–64 | nn (xx.x%) | nn (xx.x%) |
| ≥65 | nn (xx.x%) | nn (xx.x%) |
| Sex | | |
| n | nnn | nnn |
| Male | nn (xx.x%) | nn (xx.x%) |
| Female | nn (xx.x%) | nn (xx.x%) |
| Weight (kg) at baseline | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x |
| Min-max | xx-xx | xx-xx |
| Height (cm) at baseline | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x |
| Min-max | XX-XX | xx-xx |
| ECOG Category at baseline | | |
| n | nnn | nnn |
| 0 | nn (xx.x%) | nn (xx.x%) |
| >=1 | nn (xx.x%) | nn (xx.x%) |
| 9.49 | | |

- 1. Analysis population: ITT
- 2. Template ID: DMT01
- 3. Program name: T\_DM
- 4. CRF: Demographics, ECOG Performance Status, Vital Signs
- 5. See section 4.1 for identifying further variables that may be included in this output.

# 10.11 Output 11 Baseline Disease Characteristics and Prognostic Markers

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Ouration since initial diagnosis* | 10 to | \$1000 D000 D0 |
| (months) | | |
| n | nn | nn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min–max | XX-XX | xx-xx |
| Ann Arbor Stage at initial diagnosis | | |
| n | nn | nn |
| Stage 1 | nn (xx.x%) | nn (xx.x%) |
| Stage 2 | nn (xx.x%) | nn (xx.x%) |
| Stage 3 | nn (xx.x%) | nn (xx.x%) |
| Stage 4 | nn (xx.x%) | nn (xx.x%) |
| nitial FL grade** | | |
| n | nn | nn |
| Grade 1 | nn (xx.x%) | nn (xx.x%) |
| Grade 2 | nn (xx.x%) | nn (xx.x%) |
| Grade 3a | nn (xx.x%) | nn (xx.x%) |
| Ungraded | nn (xx.x%) | nn (xx.x%) |
| Ouration since diagnosis at study entry* (months) | | |
| n | nn | nn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-max | xx-xx | xx-xx |
| Ann Arbor Stage at study entry | | |
| n | nn | nn |
| Stage 1 | nn (xx.x%) | nn (xx.x%) |
| Stage 2 | nn (xx.x%) | nn (xx.x%) |
| Stage 3 | nn (xx.x%) | nn (xx.x%) |
| Stage 4 | nn (xx.x%) | nn (xx.x%) |
| FL Grade at study entry** | | |
| n | nn | nn |
| Grade 1 | nn (xx.x%) | nn (xx.x%) |
| Grade 2 | nn (xx.x%) | nn (xx.x%) |
| Grade 3a | nn (xx.x%) | nn (xx.x%) |
| Ungraded | nn (xx.x%) | nn (xx.x%) |
| Prior anti-lymphoma therapy | | |
| N | | |

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| Lines of prior anti-lymphoma<br>therapy | | |
| N | nn | nn |
| 1 | nn (xx.x%) | nn (xx.x%) |
| 2 | nn (xx.x%) | nn (xx.x%) |
| >=3 | nn (xx.x%) | nn (xx.x%) |
| Prior anti-CD20 agents | | |
| N | nn | nn |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| Prior autologous stem cell<br>transplant | | |
| N | nn | nn |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| Prior cancer radiotherapy | | |
| N | nn | nn |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| Total number of risk factors for IPI at initial Diagnosis (DLBCL)*** | | |
| N | nn | nn |
| Low (0 to 2) | nn (xx.x%) | nn (xx.x%) |
| High (3 to 5) | nn (xx.x%) | nn (xx.x%) |
| Total number of risk factors for IPI at study entry (DLBCL)*** | | |
| N | nn | nn |
| Low (0 to 2) | nn (xx.x%) | nn (xx.x%) |
| High (3 to 5) | nn (xx.x%) | nn (xx.x%) |
| Total number of risk factors for FLIPI at initial Diagnosis (FL)** | | |
| N | nn | nn |
| Low (0 or 1) | nn (xx.x%) | nn (xx.x%) |
| Intermediate (2) | nn (xx.x%) | nn (xx.x%) |
| High (3 to 5) | nn (xx.x%) | nn (xx.x%) |
| Total number of risk factors for FLIPI<br>at study entry (FL)*** | | |

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| N | nn | nn |
| Low (0 or 1) | nn (xx.x%) | nn (xx.x%) |
| Intermediate (2) | nn (xx.x%) | nn (xx.x%) |
| High (3 to 5) | nn (xx.x%) | nn (xx.x%) |
| Total number of risk factors for FLIPI2 at initial Diagnosis (FL)** | | |
| N | nn | nn |
| Low (0 or 1) | nn (xx.x%) | nn (xx.x%) |
| Intermediate (2) | nn (xx.x%) | nn (xx.x%) |
| High (3 to 5) | nn (xx.x%) | nn (xx.x%) |
| Total number of risk factors for FLIPI2 at study entry (FL)*** | | |
| N | nn | nn |
| Low (0 or 1) | nn (xx.x%) | nn (xx.x%) |
| Intermediate (2) | nn (xx.x%) | nn (xx.x%) |
| High (3 to 5) | nn (xx.x%) | nn (xx.x%) |
| B-Symptom: unexplained fever <b>greater</b> | | |
| than 38 degree C | | |
| N | nn | nn |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| B-Symptom: night sweats | | |
| N | nn | nn |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| B-Symptom: unexplained weight loss<br>greater than 10% in less than or equal<br>6 months | | |

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| N | nn | nn |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| SPD | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | xx.x |
| Min-max | xx-xx | xx-xx |
| Bulk Disease | | |
| n | nnn | nnn |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| LDH | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-max | xx-xx | xx–xx |
| Bone marrow involvement | | |
| n | nnn | nnn |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| PROTECTION OF THE PROTECTION O | | |

#### Programming notes:

- 1. Analysis population: ITT
- 2. Template ID: DMT01
- 3. Program name: T DM HIS
- 4. \*Duration since initial diagnosis: time from date of initial histological diagnosis to date of first study drug
- 5. \*Duration since diagnosis at study entry: time from date of diagnosis at study entry to date of first study drug
- 6. Generate this output for DLBCL and FL respectively (\*\*: only applicable for FL groups, \*\*\*: only applicable for DLBCL groups)
- 7. Lines of prior anti-lymphoma chemotherapy: maximum lines of anti-lymphoma therapy
- 8. CRF: NHL history, NHL prognostic factors, prior anti-lymphoma therapy, prior anti-CD20 agents, prior autologous stem cell transplant, prior anti-lymphoma radiotherapy
- 9. Further variables that may be included here are listed in section 4.2

Note: For FLIPI/IP category, follow study SMT instruction if different from the mockup.

# 10.12 Output 12 Peripheral Neuropathy History

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Patients with history of peripheral neuropathy | | , |
| n | nn | nn |
| Status of peripheral neuropathy | | |
| n | nn | nn |
| Resolved | nn (xx.x%) | nn (xx.x%) |
| Ongoing with treatment | nn (xx.x%) | nn (xx.x%) |
| Ongoing without treatment | nn (xx.x%) | nn (xx.x%) |
| Type of peripheral neuropathy | | |
| n | nn | nn |
| Sensory only | nn (xx.x%) | nn (xx.x%) |
| Motor only | nn (xx.x%) | nn (xx.x%) |
| Sensory and motor | nn (xx.x%) | nn (xx.x%) |
| Unable to determine | nn (xx.x%) | nn (xx.x%) |

- 1. Analysis population: ITT
- 2. Template ID: DMT01
- 3. Program name: T PN
- 4. CRF: Peripheral Neuropathy Medical History and Baseline Conditions
- 5. Status of PN: If a patient had more than one record, the status will be determined according to the sequence: Ongoing with treatment, ongoing without treatment, and then resolved.
- 6. Type of PN: If a patient had more than one record, the type of PN should include all the types which were presented in each record.
- 7. This output is only applied to studies with polatuzumab or lenalidomide.

# 10.13 Output 13 Medical History

| MedDRA System Organ Class<br>MedDRA Preferred Term | Treatment<br>Group 1 (N=nn) | Treatment<br>Group 2 (N=nn) |
|---|---|---|
| Total number of patients with at least one condition | nn (xx.x%) | nn (xx.x%) |
| Overall total number of conditions | nn | nn |
| VASCULAR DISORDERS | | |
| Total number of patients with at least one condition | nn (xx.x%) | nn (xx.x%) |
| HYPERTENSION | nn (xx.x%) | nn (xx.x%) |
| VARICOSE VEINS | nn (xx.x%) | nn (xx.x%) |
| ••• | | |
| Total number of conditions | nn | nn |

Investigator text for medical history conditions coded using MedDRA version xx.x. Percentages are based on N in the column headings.

#### Programming notes:

Analysis population: ITT
 Template ID: MHT01
 Program name: T\_MH

4. CRF: General Medical History and Baseline Conditions

# 10.14 Output 14 Listing of Previous Systemic Anti-lymphoma Therapy

| Center/<br>Patient ID | Age/Sex/Race | Line of<br>Therapy | Chemotherapy<br>Regimen | Chemotherapy<br>Cycles | First<br>Agent<br>Day | Last<br>Agent<br>Day | Best Response | PD | Anti-CD2O<br>Agent | Abti-CD20<br>Dose | Autologous<br>Stem Cell<br>Transplant |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1st | СНОР | 6 | | | CR | YES | Rituximab | | YES |

- 1. Analysis population: ITT
- 2. Program name: l\_cm
- 3. CRF: Prior anti-lymphoma therapy, prior anti-CD20 agents, prior autologous stem cell transplant

10.15 Output 15 Previous Systemic Anti-lymphoma Therapy

| Total number of patients with at least one treatment | Treatment<br>Group 1<br>(N=nn) | Treatment<br>Group 2<br>(N=nn) |
|---|---|---|
| Anti-lymphoma Therapy Backbone | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn |
| XXXXXXX | nn (xx.x%) | nn (xx.x%) |
| YYYYYY | nn (xx.x%) | nn (xx.x%) |
| <b>ZZZZZZZ</b> | nn (xx.x%) | nn (xx.x%) |
| Anti-CD20 as Induction Treatment | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn |
| XXXXXXX | nn (xx.x%) | nn (xx.x%) |
| YYYYYY | nn (xx.x%) | nn (xx.x%) |
| <u> </u> | nn (xx.x%) | nn (xx.x%) |
| Anti-CD20 as Induction and Maintenance<br>Treatment | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn |
| XXXXXXX | nn (xx.x%) | nn (xx.x%) |
| YYYYYY | nn (xx.x%) | nn (xx.x%) |
| 77777777 | nn (xx.x%) | nn (xx.x%) |
| Autologous Stem Cell Transplant | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn |
| Autologous Stem Cell Transplant | nn (xx.x%) | nn (xx.x%) |

Multiple uses of a specific medication for a patient were counted once in the frequency for the medication. Likewise, multiple uses within a specific medication class for a patient were counted once in the frequency for the medication class.

- 1. Analysis population: ITT
- 2. Program name: T\_PALT
- 3. CRF: Prior anti-lymphoma therapy, prior anti-CD20 agents, prior autologous stem cell transplant

## 10.16 Output 16 Response to Previous Systemic Anti-lymphoma Therapy

| | Treatment<br>Group 1<br>(N=nn) | Treatment<br>Group 2<br>(N=nn) |
|---|---|---|
| Lines of prior anti-lymphoma therapy | | |
| n | nn | nn |
| Mean (SD) | x.x (x.x) | x.x (x.x) |
| Median | x.x | x.x |
| 25 <sup>th</sup> -75th | x.x-x.x | x.x-x.x |
| Min-Max | X-X | x-x |
| Refractory to last prior anti-CD20 agents* | | |
| n | nn (xx.x%) | nn (xx.x%) |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| Refractory to last prior anti-lymphoma therapy** | | |
| n | nn (xx.x%) | nn (xx.x%) |
| Yes | nn (xx.x%) | nn (xx.x%) |
| No | nn (xx.x%) | nn (xx.x%) |
| Time from last prior anti-lymphoma therapy (days)*** | | |
| n | nn | nn |
| Mean (SD) | x.x (x.x) | x.x (x.x) |
| Median | x.x | x.x |
| 25 <sup>th</sup> -75th | x.x-x.x | x.x-x.x |
| Min-Max | x-x | x-x |

<sup>\*</sup> Defined as no response or progression on or relapse within 6 months of last antilymphoma therapy among patients whose last prior regimen contained anti-CD20

1. Analysis population: ITT

2. Program name: T PALT R

<sup>\*\*</sup> Defined as no response or progression on or relapse within 6 months of last antilymphoma therapy

<sup>\*\*\*</sup> Defined as time from end date of last anti-lymphoma therapy to first dose date Programming notes:

# 10.17 Output 17 Listing of Follow-up New Anti-lymphoma Therapy

| Center/<br>Patient ID | Age/Sex/Race | Line of<br>Therapy | Regimen | Last<br>Study<br>Dose<br>Day | First<br>Agent<br>Day | Last<br>Agent<br>Day | Anti-CD2O<br>Agent | Surgery/Procedure<br>description | Site | Surgery/Procedure<br>Day |
|---|---|---|---|---|---|---|---|---|---|---|
| | | 1st | СНОР | | | | Rituximab | | | |

- 1. Analysis population: Safety
- 2. Program name: L\_PALT
- 3. CRF: Follow-up New Anti-Lymphoma Therapy, Regimen

## 10.18 Output 18 Follow-up New Anti-lymphoma Therapy

| Total number of patients with at least one treatment | Treatment<br>Group 1<br>(N=nn) | Treatment<br>Group 2<br>(N=nn) |
|---|---|---|
| Chemotherapy | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn |
| XXXXXXX | nn (xx.x%) | nn (xx.x%) |
| YYYYYY | nn (xx.x%) | nn (xx.x%) |
| ZZZZZZZZ | nn (xx.x%) | nn (xx.x%) |
| **** | | |
| Anti-CD20 | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn |
| XXXXXXX | nn (xx.x%) | nn (xx.x%) |
| YYYYYY | nn (xx.x%) | nn (xx.x%) |
| ZZZZZZZZ | nn (xx.x%) | nn (xx.x%) |
| Autologous Stem Cell Transplant | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn |
| Autologous Stem Cell Transplant | nn (xx.x%) | nn (xx.x%) |

Multiple uses of a specific medication for a patient were counted once in the frequency for the medication. Likewise, multiple uses within a specific medication class for a patient were counted once in the frequency for the medication class.

- 1. Analysis population: Safety
- 2. Program name: T NALT
- 3. CRF: Follow-up New Anti-Lymphoma Therapy, Regimen
- 4. Provide two separate outputs if necessary: Anti-Lymphoma Treatments Administered Before Progression and Anti-Lymphoma Treatments Administered After Progression

## 10.19 Output 19 Concomitant Medication

| Class<br>Other Treatment | Treatment<br>Group 1 (N=nn) | Treatment<br>Group 2 (N=nn) |
|---|---|---|
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| Total number of treatments | nnn | nnn |
| CORTICOSTEROIDS | | |
| Total number of patients with at least one treatment | nn (xx.x%) | nn (xx.x%) |
| PREDNISONE | nn (xx.x%) | nn (xx.x%) |
| PREDNISOLONE | nn (xx.x%) | nn (xx.x%) |
| ••• | | |
| Total number of treatments | nnn | nnn |

Multiple uses of a specific medication for a patient were counted once in the frequency for the medication. Likewise, multiple uses within a specific medication class for a patient were counted once in the frequency for the medication class.

#### Programming notes:

1. Analysis population: Safety

2. Template ID: CMT01

3. Program name: T\_CM

4. CRF: Concomitant medication

5. Concomitant treatments are defined as any medication starting on or after the first day of study treatment

#### 10.20 Output 20 Previous-Concomitant Medications

#### Programming notes:

1. Analysis population: Safety

2. Template ID: CMT01

3. Program name: T PCM

4. CRF: Concomitant medication

5. Previous-Concomitant treatments are any medication started before study treatment start and ending after the start of study treatment

#### 10.21 Output 21 Previous Medications

#### Programming notes:

1. Analysis population: Safety

2. Template ID: CMT01

3. Program name: T\_PM

4. CRF: Concomitant medication

5. Previous treatments are defined as all treatments with an end date occurring before date of first study treatment.

#### 10.22 Output 22 Surgery and Procedure History

| Class<br>Other Treatment | Treatment<br>Group 1 (N=nn) | Treatment<br>Group 2 (N=nn) |
|---|---|---|
| Total number of patients with at least one surgery and procedure | nn (xx.x%) | nn (xx.x%) |
| Total number of surgery and procedure | nnn | nnn |
| Total number of patients with at least one surgery and procedure | nn (xx.x%) | nn (xx.x%) |
| XXXXXXXX | nn (xx.x%) | nn (xx.x%) |
| XXXXXXXX | nn (xx.x%) | nn (xx.x%) |
| Total number of surgery and procedure | nnn | nnn |

#### Programming notes:

1. Analysis population: Safety

2. Template ID: CMT01

3. Program name: T\_XP

4. CRF: Surgery and Procedure History

## 10.23 Output 23 Glossary of Superclass terms, Preferred Terms and Verbatim Terms for Concomitant Medications

| Medication Class | Standardized Term | Verbatim Term |
|------------------|-------------------|---------------|
| XXXXXXXXXXXX | | |
| | XXXXXXXXXXX | XXXXXXXXXXX |
| | | XXXXXXXXXXXX |
| | XXXXXXXXXXXX | XXXXXXXXXXXX |
| | XXXXXXXXXXXX | XXXXXXXXXXX |
| | XXXXXXXXXXXX | XXXXXXXXXXXX |
| | | XXXXXXXXXXXX |
| | | XXXXXXXXXXXX |
| | XXXXXXXXXXXX | XXXXXXXXXXXX |
| | | XXXXXXXXXXXX |
| | XXXXXXXXXXXX | XXXXXXXXXXX |
| XXXXXXXXXXXXX | | |
| | XXXXXXXXXXXX | XXXXXXXXXXX |
| | XXXXXXXXXXXX | XXXXXXXXXXXX |

#### Programming notes:

Template ID: AEL01
 Program name: L\_CM

3. CRF: Concomitant medication

4. Including previous, previous-concomitant, and concomitant medications

# 10.24 Output 24 Listing of Study Drug Exposure

| Center/<br>Patient ID | Age/Sex/Race | Date of First<br>Study Drug<br>Administration | Cycle | Treatment | Start Day | End Day | Dose | Unit | Reason for<br>Dose<br>Adjustment |
|---|---|---|---|---|---|---|---|---|---|
| | | | 1 | Study drug 1 | х | x | xx | xx | Adverse event |
| | | | | Study drug 2 | x | x | xx | xx | |
| | | | | Study drug 3 | x | x | xx | xx | |
| | | | n | xx | nn | nn | XX | XX | |

#### Programming notes:

1. Analysis population: Safety

2. Program name: L\_EX

3. CRF: study drug administration

4. For BO29563 and BO29561 display visit label instead of Cycle

# 10.25 Output 25 Study Drug Exposure during Induction Phase

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Study Drug 1 | | |
| Treatment duration (months) | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | xx.x |
| Min-max | XX-XX | XX-XX |
| Number of cycles | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x |
| Min-max | xx-xx | xx-xx |
| Treatment duration (Cycles) | | |
| n | nnn | nnn |
| 1–6 | nn (xx.x%) | nn (xx.x%) |
| 7-12 | nn (xx.x%) | nn (xx.x%) |
| 13-18 | nn (xx.x%) | nn (xx.x%) |
| 19-24 | nn (xx.x%) | nn (xx.x%) |
| >=25 | nn (xx.x%) | nn (xx.x%) |
| Total number of dose | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX | xx |
| Min-max | xx-xx | xx-xx |
| Total cumulative dose (mg) | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x |
| Min-max | XX-XX | xx-xx |
| Dose intensity (%) adjusted for dose modification and delay | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | xx.x |
| Min-max | xx-xx | xx-xx |
| Study Drug 2 | | |
| Study Drug 3 | | |

Treatment duration is the date of the last dose of study medication minus the date of the first dose plus 1 day.

Dose intensity (%) is the cumulative total dose actually received up to the last cycle actually received divided by the expected dose up to the last time point when any component of study medication was actually received.

#### Programming notes:

- 1. Analysis population: Safety
- 2. Template ID: EXT01
- 3. Program name: T\_EX\_IN
- 4. Treatment duration (days)=(date of last dose-date of first dose)+1
- 5. Treatment cycles: based on the actual cycles
- 6. Exposure by Cycle is optional

# **10.26 Output 26 Study Drug Exposure During Maintenance/Consolidation Phase**

- 1. Analysis population: Safety
- 2. Template ID: EXT01
- 3. Program name: T EX MC
- 4. Treatment duration (days)=(date of last dose-date of first dose)+1
- 5. Treatment cycles: based on the actual cycles
- 6. Exposure by Cycle is optional.

# 10.27 Output 27 Glossary of Adverse Event Preferred Terms and Investigator-Specified Terms

| MedDRA System Organ Class | MedDRA Preferred Term | Investigator-Specified Adverse Event Term |
|---|---|---|
| BLOOD AND LYMPHATIC SYSTEM | | |
| DISORDERS | ANAEMIA NOS | ANAEMIA |
| | | ANEMIA |
| | LEUCOCYTOSIS NOS | LEUKOCYTOSIS |
| | LEUCOPENIA NOS | LEUKOPENIA |
| | LYMPHADENOPATHY | NECROTIC LYMPH NODE |
| | | SWOLLEN GLANDS IN THROAT |
| | | SWOLLEN THROAT GLANDS |
| | FEBRILE NEUTROPENIA | FEBRILE NEUTROPENIA |
| | | NEUTROPENIC FEVER |
| | NEUTROPENIA | NEUTROPENIA |
| CARDIAC DISORDERS | | |
| | CARDIOMYOPATHY NOS | CARDIOMYOPATHY |
| | CONGESTIVE (DILATED) CARDIOMYOPATHY | DILATED CARDIOMYOPATHY |
| | ANGINA PECTORIS | ANGINA PECTORIS |

## Programming notes:

Template ID: AEL01
 Program name: L\_AE\_PT

#### 10.28 Output 28 Listing of Adverse Events

| Center/Patient ID-<br>Age/Sex/Race<br>MedDRA Preferred Term | Date of First<br>Study Drug<br>Administration | Study Day<br>of Onset | AE<br>Duration<br>in Days | Most<br>Extreme<br>CTC<br>Grade | Outcome<br>(1) | Treatment<br>for AE | Relation to<br>Study drug | Action with<br>Study drug<br>(2) | Reason<br>Classified<br>as Serious<br>(3) |
|---|---|---|---|---|---|---|---|---|---|
| nnnnnn/nnnnn-nn/x/x xxxxxxxxxxx | nnxxxnnnn | nn | 12 | 4 | 2 | xxx | A:No, G:No,<br>V:Yes | A:3, G:2, V:3 | n |

<sup>\*:</sup> SAE (1) Outcome: 1 = fatal; 2 = not recovered/not resolved; 3 = recovered/resolved; 4 = recovered/resolved with sequelae;

- (2) Action taken with study drug: 1 = dose not changed; 2 = dose reduced; 3 = drug interrupted; 4 = drug withdrawn;
- 5 = not applicable; 6 = unknown.
- (3) Reason classified as serious: 1 = resulted in death; 2 = life threatening; 3 = required prolonged in patient hospitalization;

4= disabling; 5= a congenital anomaly/birth defect in offspring of study subject; 6= does not meet any of the above serious

criteria, but may jeopardize the subject, and may require medical or surgical intervention to prevent one of the outcomes listed

above.

Relation to Study Drug & Action with Study drug: A = Atezolizumab; G = GA101; V = Venetoclax;

#### Programming notes:

1. Analysis population: Safety

2. Template ID: AEL02

3. Program name: L\_AE

4. The final footnote is dependent on which study drugs are given

<sup>5 =</sup> recovering/resolving; 6 = unknown.

## 10.29 Output 29 Listing of Serious Adverse Events

#### Programming notes:

1. Analysis population: Safety

Template ID: AEL02
 Program name: L\_AES

### 10.30 Output 30 Listing of Grade 3, 4, 5 Adverse Events

#### Programming notes:

1. Analysis population: Safety

Template ID: AEL02
 Program name: L\_AE345

# 10.31 Output 31 Listing of Adverse Events Leading to Discontinuation of Any Study Drug

#### Programming notes:

1. Analysis population: Safety

Template ID: AEL02
 Program name: L\_AEW

# 10.32 Output 32 Listing of Adverse Events Leading to Dose Modification or Interruption of Any Study Drug

#### Programming notes:

1. Analysis population: Safety

Template ID: AEL02
 Program name: L\_AEM

## 10.33 Output 33 Listing of Adverse Events Leading to Death

#### Programming notes:

1. Analysis population: Safety

Template ID: AEL02
 Program name: L\_AED

#### 10.34 Output 34 Listing of Potential Adverse Events of Special Interest

Programming notes:

1. Analysis population: Safety

Template ID: AEL02
 Program name: L\_AESI

4. Definition: see Table in 6.2.2 Selected AEs and Potential AE of Special Interest

Note: For BO29561-3 an additional listing based on AESI ticked on eCRF AESI page will be created. AESI will be summarized by tickbox categories. Only AESI with causality to Atezo suspected and onset >= cycle 2 start will be included.

## 10.35 Output 35 Listing of Selected Adverse Events

Programming notes:

1. Analysis population: Safety

Template ID: AEL02
 Program name: L AESE

4. Definition of selected AE (see table in section 6.2.2)

Note: listing 34 and 35 may be combined depending on individual studies. The title becomes "Listing of Adverse Events of Selected and Special Interest"

#### 10.36 Output 36 Safety Summary

| | Treatment Group 1 (N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Total number of AEs | nn | nn |
| Total number of patients with at least one | | |
| AE | nn (xx.x%) | nn (xx.x%) |
| Grade 5 AE | nn (xx.x%) | nn (xx.x%) |
| Grade 3-5 AE | nn (xx.x%) | nn (xx.x%) |
| Serious AE | nn (xx.x%) | nn (xx.x%) |
| AE leading to any study treatment discontinuation AE leading to dose reductions AE leading to drug interruptions | nn (xx.x%) | nn (xx.x%) |
| AE leading to study discontinuation | nn (xx.x%) | nn (xx.x%) |
| Related to Drug 1 AE | nn (xx.x%) | nn (xx.x%) |
| Related to Drug 1 Grade 3-5AE | nn (xx.x%) | nn (xx.x%) |
| Related to Drug 1 SAE | nn (xx.x%) | nn (xx.x%) |
| Related to Drug 2 AE | nn (xx.x%) | nn (xx.x%) |
| Related to Drug 2 Grade 3-5 AE | nn (xx.x%) | nn (xx.x%) |
| Related to Drug 2 SAE | nn (xx.x%) | nn (xx.x%) |
| Related AE (to at least one treatment) leading to study treatment discontinuation (of all treatments) | nn (xx.x%) | nn (xx.x%) |
| Related AE (to at least one treatment) leading to study discontinuation | nn (xx.x%) | nn (xx.x%) |

Investigator text for AEs encoded using MedDRA version xx.x. Percentages are based on N in the column headings. Includes AEs with onset from first dose of study drug through XX days after last dose of study drug

- 1. Analysis population: Safety
- 2. Template ID: AET01
- 3. Program name: T AE OSAFE
- 4. Reporting period: All adverse events will be reported until XX days (study specific) after the last dose of study treatment. An exception is Grade 3 and 4 infections (both related and unrelated), which should be reported until up to 2 years after the last dose of study treatment. Study BO29562: An exception is secondary malignancies (both related and unrelated), which should be reported until up to 6months after the last dose of lenalidomide.
- 5. All the following safety outputs will be produced by study phase

# 10.37 Output 37 Adverse Events

| MedDRA System Organ Class<br>MedDRA Preferred Term | Treatment Group<br>1 (N=nn) | Treatment Group<br>2 (N=nn) |
|---|---|---|
| Total number of patients with at least one AE | nn (xx.x%) | nn (xx.x%) |
| Overall total number of AEs | nn | nn |
| SOC 1 | | |
| Total number of patients with at least one AE event | nn (xx.x%) | nn (xx.x%) |
| PT1 | nn (xx.x%) | nn (xx.x%) |
| PT2 | nn (xx.x%) | nn (xx.x%) |
| PT3 | nn (xx.x%) | nn (xx.x%) |
| PT4 | nn (xx.x%) | nn (xx.x%) |
| Total number of events | nn | nn |
| SOC 2 | | |
| Total number of patients with at least one AE | nn (xx.x%) | nn (xx.x%) |
| PT1 | nn (xx.x%) | nn (xx.x%) |
| PT2 | nn (xx.x%) | nn (xx.x%) |
| PT3 | nn (xx.x%) | nn (xx.x%) |
| PT4 | nn (xx.x%) | nn (xx.x%) |
| Total number of events | nn | nn |
| ••• | | |

Investigator text for AEs encoded using MedDRA version xx.x. Percentages are based on N in the column headings. Includes AEs with onset from first dose of study drug through xx days after last dose of study drug

Programming notes:

1. Analysis population: Safety

Template ID: AET02
 Program name: T\_AE

#### 10.38 Output 38 Grade 3, 4, 5 Adverse Events

Programing notes:

1. Analysis population: Safety

Template ID: AET02
 Program name: T\_AE345

#### 10.39 Output 39 Serious Adverse Events

Programing notes:

1. Analysis population: Safety

Template ID: AET02
 Program name: T\_AES

# 10.40 Output 40 Adverse Events Leading to Discontinuation of Any Study Drug

Programing notes:

1. Analysis population: Safety

Template ID: AET02
 Program name: T\_AEW

#### 10.41 Output 41 Potential Adverse Events of Special Interest

Programing notes:

1. Analysis population: Safety

2. Template ID: AET02

3. Program name: T\_AESPECIAL

4. Summarized by AESI category (see table 6.2.2)

Note: "Adverse events of special interest" may be combined with "Selected Adverse Events".

Note: For BO29561-3 an additional summary based on AESI ticked on eCRF AESI page will be created. AESI will be summarized by tickbox categories. Only AESI with causality to Atezo suspected and onset >= cycle 2 will be included.

### 10.42 Output 42 Selected Adverse Events

Programing notes:

1. Analysis population: Safety

2. Template ID: AET02

3. Program name: T\_AESELECT

4. Summarized by AESI category (SMQ) and Preferred Term

Note: "Adverse events of special interest" may be combined with "Selected Adverse Events".

10.43 Output 43 Categorical Summary of Adverse Events of Special Interest

| | Treatment Group 1 |
|---|---|
| | <del>(N - xx)</del> |
| No. of patients with at least one AE | <del>xx (xx %)</del> |
| No. of patients with grade 1 AEs | <del>xx (xx %)</del> |
| No. of patients with grade 2 AEs | <del>xx (xx %)</del> |
| No. of patients with grade 3 AEs | <del>xx (xx %)</del> |
| No. of patients with grade 4 AEs | <del>xx (xx %)</del> |
| No. of patients with grade 5 AEs | <del>xx (xx %)</del> |
| No. of patients with missing grade-AEs | <del>хх (хх %)</del> |
| No. of patients with serious AE | <del>xx (xx %)</del> |
| Tetal Ne. of AEs | <del>xx</del> |
| No. of grade 1 AEs | ×× |
| No. of grado 2 AEs | <del>XX</del> |
| No. of grade 3 AEs | <del>XX</del> |
| No. of grade 4 AEs | <del>XX</del> |
| No. of grade 15 AEs | <del>xx</del> |
| No. of AEs with missing grade | <del>XX</del> |
| No. of serious AEs | <del>××</del> |
| No. of AEs with missing seriousness | <del>)(X</del> |
| Tetal No. of patients with at least one AE: | <del>XX</del> |
| No. of patients with ant body dose interrupted due to AE | <del>xx (xx %)</del> |
| No. of patients with ant body withdrawn due to AE | <del>хх (хх %)</del> |
| No. of patients with atezolizumab interrupted due to AE | <del>xx (xx %)</del> |
| No. of patients with atezolizumab withdrawn due to AE | <del>xx (xx %)</del><br><del>xx (xx %)</del> |
| No. of patients with chemotherapy dose reduced due to AE | ** (** %) |
| No. of patients with chemotherapy interrupted due to AE | <del>xx (xx %)</del> |
| No. of patients with chemotherapy withdrawn due to AE | <del>xx (xx %)</del> |
| 1 | <del>хх (хх %)</del> |
| No. of patients with any treatment dose reduced due to AE | <del>xx (xx %)</del> |
| No. of patients with any treatment interrupted due to AE | <del>xx (xx %)</del> |
| No. of patients with any treatment withdrawn due to AE | ** (** %) |
| No. of patients with at least one AE unresolved or engoing | ** (** %) |
| No. of patients with treatment received for AE | <del>xx (xx %)</del> |
| No. of patients without treatment received for AE | <del>xx (xx %)</del> |

Percentages are based on the number of patients with at least one AE (except the first-block of the output where the percentages are based on N).

When calculating the number of patients with AEs of a specific grade only the highest AE grade per patient is taken into account.

All occurrences of the same adverse event in one patient are counted separately. Investigator text for AEs encoded using MedDRA vxx.x.

- 1. Analysis population: Safety
- 2. Program name: T\_AE\_C\_AESPECIAL
- 3.—Definition: see Table in 6.2.2 Selected AEs and Potential AE of Special Interest
- 4.—'Chemotherapy' can be replaced by the actual study chemotherapy term, e.g. Bendamustine

#### 10.44 Output 44 Categorical Summary of Selected Adverse Events

#### **Programing notes:**

- 1. Analysis population: Safety
- 2.—Program name: T AE C AESELECT
- 3.—Definition: see Table in 6.2.2 Selected AEs and Potential AE of Special Interest

#### 10.45 Output 45 Adverse Events by Cycle

| Treatment Cycles | Treatment Group 1 |
|--------------------------------------------------|-------------------|
| | (N = xx) |
| Cycle 1 | |
| Patients with at least one AE | xx (xx%) |
| Number of AEs | XX |
| Number of grade 3-4 AEs | XX |
| Number of fatal AEs | XX |
| Number of serious AEs | XX |
| Number of AEs leading to ant body withdrawal | XX |
| Number of AEs leading to atezolizumab withdrawal | XX |
| Number of AEs leading to chemotherapy withdrawal | XX |
| n | XX |
| Cycle 2 | |
| Patients with at least one AE | xx (xx%) |
| Number of AEs | XX |
| Number of grade 3-4 AEs | XX |
| Number of fatal AEs | XX |
| Number of serious AEs | XX |
| Number of AEs leading to ant body withdrawal | XX |
| Number of AEs leading to atezolizumab withdrawal | XX |
| Number of AEs leading to chemotherapy withdrawal | XX |
| n | XX |
| Cycle x | |

Investigator text for AEs encoded using MedDRA vxx.x.

n is a number of patients received study drug at each cycle.

Percentages are based on n.

Multiple occurrences of the same adverse event in one individual counted only once for each cycle.

#### Programing notes:

- 1. Analysis population: Safety
- 2. Program name: T\_AE\_C\_AECYC
- 3. 'Chemotherapy' can be replaced by the actual study chemotherapy term, e.g. Bendamustine

#### 10.46 Output 46 Potential Adverse Events of Special Interest by Cycle

1. Analysis population: Safety

2. Program name: T AESI C AECYC

3. 'Chemotherapy' can be replaced by the actual study chemotherapy term, e.g. Bendamustine

#### 10.47 Output 47 Selected Adverse Events by Cycle

Programing notes:

1. Analysis population: Safety

2. Program name: T\_AESE\_C\_AECYC

3. 'Chemotherapy' can be replaced by the actual study chemotherapy term, e.g. Bendamustine

#### 10.48 Output 48 Adverse Events by Highest NCI CTCAE Grade

| MedDRA System Organ Class and<br>Preferred Term | Grade | Treatment<br>Group 1 (N=nn) | Treatment<br>Group 2 (N=nn) |
|---|---|---|---|
| | -Any Grade- | nn | nn |
| | 1 | nn | nn |
| | 2 | nn | nn |
| | 3 | nn | nn |
| | 4 | nn | nn |
| | 5 | nn | nn |
| BLOOD AND LYMPHATIC SYSTEM DISORDERS | | | |
| - Overall - | -Any Grade- | nn | nn |
| | 1 | nn | nn |
| | 2 | nn | nn |
| | 3 | nn | nn |
| | 4 | nn | nn |
| | 5 | nn | nn |
| NEUTROPENIA | -Any Grade- | nn | nn |
| | 1 | nn | nn |
| | 2 | nn | nn |
| | 3 | nn | nn |
| | 4 | nn | nn |
| | 5 | nn | nn |

Investigator text for AEs encoded using MedDRA version xx.x. Multiple occurrences of the same AE in one individual are counted once at the maximum intensity for this term. The Any Intensity rows present the number of AEs reported at any intensity across all patients. Patients experiencing > 1 event (different PTs) within a SOC will have all unique events contributing to this count. Includes AEs with onset from first dose of study drug through xx days after last dose of study drug

#### Programing notes:

1. Analysis population: Safety

2. Template ID: AET04

3. Program name: T\_AE\_CTC
# 10.49 Output 49 Most Common Adverse Event with Incidence $\geq$ 5% by Preferred Term

Programing notes:

1. Analysis population: Safety

2. Template ID: AET08

3. Program name: T\_AE\_PT\_P5

4. Display only by preferred term, not by SOC

# 10.50 Output 50 Most Common Grade 3, 4, 5 Adverse Event with Incidence $\geq$ 5% by Preferred Term

Programing notes:

1. Analysis population: Safety

2. Template ID: AET08

3. Program name: T\_AE345\_PT\_P5

# 10.51 Output 51 Duration from First Study Treatment Date to Onset of Peripheral Neuropathy

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Duration from first study treatment to onset of PN (months) | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-max | XX-XX | XX-XX |
| Duration from first study treatment to onset of grade 2 or higher PN (months) | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x |
| Min-max | XX-XX | XX-XX |

## Programing notes:

1. Analysis population: Safety

2. Template ID: NA

3. Program name: T\_DUR\_PN4. Use univariate variable analysis

5. This output is applied to studies with polatuzumab

# 10.52 Output 52 Listing of Deaths

| Center/<br>Patient ID | Age/Sex/Race | Date of First<br>Study Drug<br>Administration | Day of Last<br>Study Drug<br>Administration | Day<br>of<br>Death | Associated<br>SAE<br>Preferred<br>Term | Autopsy<br>Performed? | Cause<br>of<br>Death |
|---|---|---|---|---|---|---|---|
| | | | 12 | 62 | Myocardial<br>infarction | Yes | xxxxx |
| | | | 36 | 37 | Ischemic<br>Stroke | No | xxxxx |

## Programming notes:

1. Analysis population: Safety

2. Template ID: AEL04

3. Program name: L\_DD

# 10.53 Output 53 Deaths

| | Treatment Group<br>1 (N=nn) | Treatment Group<br>2 (N=nn) |
|---|---|---|
| All deaths | xx (xx.x%) | xx (xx.x%) |
| Adverse Events | xx (xx.x%) | xx (xx.x%) |
| Disease Progression | xx (xx.x%) | xx (xx.x%) |
| No. of deaths during treatment | | |
| Cause of death | | |
| Adverse Events | xx (xx.x%) | xx (xx.x%) |
| Disease Progression | xx (xx.x%) | xx (xx.x%) |
| No. of deaths during follow up | | |
| Cause of death | | |
| Adverse Events | xx (xx.x%) | xx (xx.x%) |
| Disease Progression | xx (xx.x%) | xx (xx.x%) |
| No. of deaths during survival follow up | | |
| Cause of death | | |
| Adverse Events | xx (xx.x%) | xx (xx.x%) |
| Disease Progression | xx (xx.x%) | xx (xx.x%) |

Deaths during the treatment are those occurred within 28 days after last study drug.

## Programming notes:

1. Analysis population: ITT

2. Program name: T\_DD

3. CRF: AE and Study Completion/Early Discontinuation

# 10.54 Output 54 Laboratory Test Results Shift Table - Highest NCI CTCAE Grade Post-Baseline

| Hemoglobin<br>g/L (Low) | | Status at Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | From | 0 | 1 | 2 | 3 | 4 | Total | Missing |
| То | | | | | | | | |
| 0 | | 13(xx%) | 0 (xx%) | 1(xx%) | 0 | 0 | 14 | 0 |
| 1 | | 58(xx%) | 63(xx%) | 4(xx%) | 0 | 0 | 125 | 0 |
| 2 | | 39(xx%) | 105(xx%) | 28(xx%) | 0 | 0 | 172 | 0 |
| 3 | | 14(xx%) | 23(xx%) | 13(xx%) | 0 | 0 | 50 | 0 |
| 4 | | 3(xx%) | 5(xx%) | 0(xx%) | 0 | 0 | 8 | 0 |
| Total | | 127(100%) | 196(100%) | 46(100%) | 0 | 0 | 360 | 0 |
| Missing | | 6 | 6 | 0 | 0 | 0 | 12 | 0 |

NCI CTCAE = National Cancer Institute Common Terminology Criteria for Adverse Events.

"n" denotes the number of patients with baseline and post-baseline lab data within this time interval. For a patient with multiple post-baseline lab abnormalities, the highest (worst) grade of these abnormalities for the given lab test is reported.

#### Programing notes:

1. Analysis population: Safety

2. Template ID: LBT14

3. Program name: T\_LB\_SHIFT

4. Use EXT\_NCICTC4 for NCI-CTCAE Grades

5. Include all hematology and chemistry lab parameters split into 2 separate outputs.

10.55 Output 55 Neutrophil Count Recovery

| | Treatment<br>Group 1 (N=nn) | Treatment Group 2 (N=nn) |
|---|---|---|
| ANC <1.0 × 109/L at EOT/EOI* | | |
| Yes | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) |
| n | XXX | XXX |
| ANC Recovery** within 3 months of follow up | | |
| Yes | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) |
| n | XXX | xxx |
| ANC Recovery** within 6 to 9 months of follow up | | |
| Yes | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) |
| n | XXX | xxx |
| ANC Recovery** within 9 to 12 months of follow up | | |
| Yes | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) |
| n | XXX | xxx |
| A ANC Recovery** after 12 months of | | |
| follow up<br>Yes | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) |
| n | xxx | xxx |

<sup>\*\*</sup> Neutrophil recovery is defined as ANC  $\geq$  1.0  $\times$  109/L, given ANC was collected after the patient received his last dose of antibody, and ANC < 1.0  $\times$  109/L the last previous visit before EOT/EOI. Where no ANC value occurs at the last drug intake, the next valid ANC assessment was taken.

Percentages are based on the number of patients with ANC <  $1.0 \times 10^9$ /L at the last previous visit before EOT/EOI.

#### Programing notes:

Analysis population: Safety
 Program name: T\_LB\_ANC

# 10.56 Output 56 Vital Signs Change from Baseline by Visit

| | | Group 1<br>(N=nnn) |
|-----------|----------------|-------------------------|
| Visit | Value at Visit | Change from<br>Baseline |
| Baseline | | |
| n | nnn | |
| Mean (SD) | xx.x (xx.x) | |
| Median | XX.X | |
| Min-max | xx.x –xx.x | |
| Cycle X | | |
| n | nnn | nnn |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | XX.X |
| Min-max | xx.x-xx.x | xx.x-xx.x |

## Programing notes:

1. Analysis population: Safety

2. Template ID: VST01

3. Program name: T\_VS\_CB

4. Analysis variables: Weight, Temperature, Respiratory rate, Pulse, SBP, DBP

# 10.57 Output 57 ECG Results Shift Table

Treatment x (N=xx)

| | Shift FROM: Baseline | | | |
|---|---|---|---|---|
| Shift TO: ECG Result at Visit | Abnormal, clinically significant | | Normal | Total |
| END OF INDUCTION COMPLETION / DISCONTINUATION | | | | |
| Abnormal, clinically significant | 0 | 0 | 0 | 0 |
| Abnormal, not clinically significant | 0 | xx (xx.xx%) | xx (xx.xx%) | xx (xx.x%) |
| Normal | 0 | xx (xx.xx%) | xx (xx.xx%) | xx (xx.xx%) |
| Total | 0 | xx (xx.xx%) | xx (xx.xx%) | xx (xx.xx%) |
| END OF MAINTENANCE COMPLETION / DISCONTINUATION | | | | |
| Abnormal, clinically significant | 0 | 0 | 0 | 0 |
| Abnormal, not clinically significant | 0 | xx (xx.xx%) | 0 | xx (xx.xx%) |
| Normal | 0 | 0 | 0 | 0 |
| Total | 0 | xx (xx.xx%) | 0 | xx (xx.xx%) |

Baseline assessment is the last valid assessment in the 28 day window before first administration of a study treatment component.

Programing notes:

1. Analysis population: Safety

2. Template ID: EGT01

3. Program name: T\_EG\_CB

4. Analysis variables: Electrocardiogram (ECG)

# 10.58 OUTPUT 58 Listing of Time-to-Event Endpoints

| Treatment group | CRTN/Pt No. | Overall Survival<br>(months) | PFS<br>(months) | EFS<br>(months) | DFS<br>(months) | Duration of<br>Response<br>(months) |
|---|---|---|---|---|---|---|
| | xxxx/xxxx | xxx | xxx | xxx | xxx | xxx |
| | | xxx | xxx* | xxx* | xxx* | |
| | | xxx | XXX | xxx | xxx | |
| | | xxx | xxx* | xxx* | xxx* | |
| | | xxx | xxx | xxx | xxx | |
| | | xxx | xxx* | xxx* | xxx* | |
| | | xxx | xxx | xxx | xxx | |

<sup>\*</sup> Censored Observation

## Programming Note:

1. Analysis population: Safety

2. Program name: L\_EF\_TTE

3. Time-to-Event endpoints are consist of overall survival, EFS, PFS, and duration of response.

## 10.59 Output 59 Listing of Tumor Response Assessment

| CRTN/PT<br>No. | Cycle | Study Day# | New<br>Lesion | Objective<br>evidence of<br>clinical<br>progression | Response not<br>including PET<br>scan results<br>(IRC) | Response based<br>upon PET-CT<br>scans (IRC) | Response not including PET scan results (Investigator) | Response based<br>upon PET-CT<br>scans<br>(Investigator) |
|---|---|---|---|---|---|---|---|---|
| xxxx/xxxx | | <del> </del> | Yes | Yes | • | , | | * |

Response will be determined on the basis of PET-CT scans or CT scans alone, using the modified Lugano 2014 criteria

#: Days from first dose of study medication

#### **Programming Note:**

- 1. Analysis population: Safety
- 2. Program name: L EF CONCORD
- 3. CRF: NHL response assessment and IRC data
- 4. Response based upon PET-CT scans include 2 results: using Lugano 2014 criteria and modified Lugano 2014 criteria (follow protocol).
- 5. Study BO29563: response assessment is also using Cheson 2007 criteria.

Note: It is ok to split the table into two: one for investigator and the other for IRC.

# 10.60 Output 60 CR Rate at End of Induction

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Based on Modified LUGANO 2014 - PET-CT | | |
| As Determined by the IRC | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% CI for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| As Determined by the Investigator | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on LUGANO 2014 - PET | | |
| As Determined by the IRC | | |
| Complete Response (CR) | xxx (xx.x %) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| As Determined by the Investigator | | |
| Complete Response (CR) | xxx (xx.x %) | xxx (xx.x %) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on Modified CHESON 2007 - CT or MRI | | |
| As Determined by the IRC | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| As Determined by the Investigator | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on Modified CHESON 2007 - CT or MRI and | J PET | |
| As Determined by the IRC | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| As Determined by the Investigator | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | (xx.x, xx.x) | ( xx.x, xx.x) |

90% Cl for rates were constructed using Clopper-Pearson method.

- 1. Analysis population: Safety
- 2. Template ID: RSPT01
- 3. Program name: T\_CRR
- 4. EOI time window: TBD
- 5. Some studies may require CR tabulation based on Cheson criteria, Lugana, or modified Lugano, follow SMT instruction.

10.61 Output 61 OR Rate at End of Induction

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Based on Modified LUGANO 2014 - PET-CT | | |
| As Determined by the IRC | | |
| Objective Response (CR, PR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% CI for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| As Determined by the Investigator | | |
| Objective Response (CR, PR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on LUGANO 2014 – PET | | |
| As Determined by the IRC | | |
| Objective Response (CR, PR) | xxx (xx.x%) | xxx (xx.x %) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| As Determined by the Investigator | | |
| Objective Response (CR, PR) | xxx (xx.x %) | xxx (xx.x %) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on Modified CHESON 2007 - CT or MRI | | |
| As Determined by the IRC | | |
| Objective Response (CR, PR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| As Determined by the Investigator | | |
| Objective Response (CR, PR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on Modified CHESON 2007 - CT or MRI and As Determined by the IRC | d PET | |
| Objective Response (CR, PR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | (xx.x, xx.x) | ( xx.x, xx.x) |
| As Determined by the Investigator | | |
| Objective Response (CR, PR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | (xx.x, xx.x) |

90% Cl for rates were constructed using Clopper-Pearson method.

- 1. Analysis population: Safety
- 2. Template ID: RSPT01

- 3. Program name: T\_ORR
- 4. EOI time window: TBD

10.62 Output 62 CR Rate at 12 Months after Initiation of Induction

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Based on PET-CT as Determined by the IRC using Lugano 2014 Criteria | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on PET-CT as Determined by the Investigator using Lugano 2014 Criteria | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on PET-CT as Determined by the IRC using modified Lugano 2014 Criteria | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on PET-CT as Determined by the Investigator using modified Lugano 2014 Criteria | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on CT alone as Determined by the IRC | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |
| Based on CT alone as Determined by the Investigator | | |
| Complete Response (CR) | xxx (xx.x%) | xxx (xx.x%) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |

90% Cl for rates were constructed using Clopper-Pearson method.

- 1. Analysis population: Safety
- 2. Template ID: RSPT01
- 3. Program name: T\_CRR12
- 4. Patient subset: Patients who have positive PET scans (CR/PR) at EOI

# 10.63 Output 63 Best Overall Response Rate

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Based on CT as Determined by the Investigator | | |
| Best Overall Response (BOR) | xxx (xx.x %) | xxx (xx.x %) |
| CR | xxx (xx.x %) | xxx (xx.x %) |
| PR | xxx (xx.x %) | xxx (xx.x %) |
| 90% Cl for Response Rates | ( xx.x, xx.x) | ( xx.x, xx.x) |

90% Cl for rates were constructed using Clopper-Pearson method.

## Programming Note:

1. Analysis population: Safety

2. Template ID: RSPT01

3. Program name: T\_BORR

10.64 Output 64 Concordance Analysis Between the IRC Determined and the Investigator Determined CR Status

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Based on PET-CT using Lugano 2014 Criteria | | |
| Number of patients evaluable for concordance | nn | nn |
| CR occurrence | | |
| Concordance | xxx (xx.x %) | xxx (xx.x %) |
| CR per investigator and CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| No CR per investigator and no CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| Discordance | xxx (xx.x %) | xxx (xx.x %) |
| CR per investigator and no CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| No CR per investigator and CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| Based on PET-CT using modified Lugano 2014<br>Criteria | | |
| Number of patients evaluable for concordance | nn | nn |
| CR occurrence | | |
| Concordance | xxx (xx.x %) | xxx (xx.x %) |
| CR per investigator and CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| No CR per investigator and no CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| Discordance | xxx (xx.x %) | xxx (xx.x%) |
| CR per investigator and no CR per IRC | xxx (xx.x %) | xxx (xx.x%) |
| No CR per investigator and CR per IRC | xxx (xx.x %) | xxx (xx.x%) |
| Based on CT alone | | |
| Number of patients evaluable for concordance CR occurrence | nn | nn |
| Concordance | xxx (xx.x %) | xxx (xx.x%) |
| CR per investigator and CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| No CR per investigator and no CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| Discordance | xxx (xx.x %) | xxx (xx.x %) |
| CR per investigator and no CR per IRC | xxx (xx.x %) | xxx (xx.x %) |
| No CR per investigator and CR per IRC | xxx (xx.x %) | xxx (xx.x %) |

## Programming Note:

1. Analysis population: Safety

2. Template ID: IRCT01

3. Program name: T\_EF\_CONCORD\_CR

## 10.65 Output 65 Duration of Response

| | Treatment Group 1<br>(N=nn) | Treatment Group 2<br>(N=nn) |
|---|---|---|
| Patients with event (%) | xxx ( xx.x %) | xxx (xx.x %) |
| PD | xxx | XXX |
| Death | xxx | XXX |
| Patients without event (%)# | xxx ( xx.x %) | xxx (xx.x %) |
| Time to event (month) | | |
| Median | xxx.x | XXX.X |
| 95% CI | (xxx, xxx) | (xxx, xxx) |
| 25% and 75%-ile | xxx, xxx | XXX, XXX |
| Range## | xxx to xxx# | xxx to xxx# |

<sup>#</sup> Censored value, ## Including censored observations

Summaries of <Time-to-Event Endpoint> (median, percentiles) are Kaplan-Meier estimates. 95% CI for median was computed using the method of Brookmeyer and Crowley.

- 1. Analysis population: Safety
- 2. Template ID: TTET01
- 3. Program name: T\_DOR
- 4. Based on CT assessment as determined by the investigators
- 5. Patient subset: Patients who have CR or PR

# 10.66 Output 66 Kaplan-Meier Curve of Duration of Response



- 1. Analysis population: Safety
- 2. Template ID: KMG01
- 3. Program name: G\_KM\_DOR
- 4. Based on CT assessment as determined by the investigators

## 10.67 Output 67 Waterfall Plot of Best Change from Baseline (%) in Indicator Lesion Size



- 1. Analysis population: Safety
- 2. Program name: G\_EF\_WTF
- 3. Based on CT assessment as determined by the investigators

## 10.68 Output 68 Spider Plot of Change from Baseline (%) in Indicator Lesion Size over Time



- 1. Analysis population: Safety
- 2. Program name: G\_EF\_SPIDER
- 3. Based on CT assessment as determined by the investigators

## 10.69 Output 69 Swimmer Plot of Time to Response and Duration of Response



- 1. Analysis population: Safety
- Program name: G\_EF\_SWIM
   Based on Lugano 2014 PET-CT assessment as determined by the investigators
- 4. Details: TBD

## 10.70 Output 70 Progression-Free Survival

| | Treatment Group 1<br>(N=nn) | Treatment Group 2 (N=nn) |
|---|---|---|
| Patients with event (%) | xxx ( xx.x %) | xxx (xx.x %) |
| PD | xxx | XXX |
| Death | xxx | XXX |
| Patients without event (%)# | xxx ( xx.x %) | xxx (xx.x %) |
| Time to event (month) | | |
| Median | xxx.x | XXX.X |
| 95% CI | (xxx, xxx) | (xxx, xxx) |
| 25% and 75%-ile | xxx, xxx | XXX, XXX |
| Range## | xxx to xxx# | xxx to xxx# |
| Time Point Analysis | | |
| 6 months duration | | |
| Patients remaining at risk | XX | XX |
| Event free rate (%) | xx.x | XX.X |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |

<sup>#</sup> Censored value, ## Including censored observations

Summaries of <Time-to-Event Endpoint> (median, percentiles) are Kaplan-Meier estimates. 95% Cl for median was computed using the method of Brookmeyer and Crowley. 95% Cl for landmark estimate was computed using Greenwood method.

#### Programming Note:

- 1. Analysis population: Safety
- 2. Program name: T EF TTE PFS
- 3. Based on CT assessment as determined by the investigators
- 4. Landmark estimates of the proportion of patients who are event free at 6 months, 9 months, 1 year, and 2 years will be provided, along with 95% asymptotic Cis using Greenwood's formula for standard errors.

### 10.71 Output 71 Kaplan-Meier Curve of Progression-free Survival

- 1. Analysis population: Safety
- 2. Program name: G\_EF\_KM\_PFS
- 3. Based on CT assessment as determined by the investigators

### 10.72 Output 72 Event-Free Survival

#### **Programming Note:**

- 1. Analysis population: Safety
- 2. Program name: T\_EF\_TTE\_EFS
- 3. Based on CT assessment as determined by the investigators
- 4. Landmark estimates of the proportion of patients who are event free at 6 months, 9 months, 1 year, and 2 years will be provided, along with 95% asymptotic Cls using Greenwood's formula for standard errors.

### 10.73 Output 73 Kaplan-Meier Curve of Event-Fee Survival

#### Programming Note:

- 1. Analysis population: Safety
- 2. Program name: G\_EF\_KM\_EFS
- 3. Based on CT assessment as determined by the investigators

## 10.74 Output 74 Disease-Free Survival

#### Programming Note:

- 1. Analysis population: Safety
- 2. Program name: T\_EF\_TTE\_DFS
- 3. Based on CT assessment as determined by the investigators
- 4. Landmark estimates of the proportion of patients who are event free at 6 months, 9 months, 1 year, and 2 years will be provided, along with 95% asymptotic Cis using Greenwood's formula for standard errors.

## 10.75 Output 75 Kaplan-Meier Curve of Disease-Fee Survival

- 1. Analysis population: Safety
- 2. Program name: G\_EF\_KM\_DFS
- 3. Based on CT assessment as determined by the investigators

## 10.76 Output 76 Overall Survival

Programming Note:

1. Analysis population: Safety

2. Program name: T\_EF\_TTE\_OS

3. Landmark estimates of the proportion of patients who are event free at 6 months, 9 months, 1 year, and 2 years will be provided, along with 95% asymptotic CIs using Greenwood's formula for standard errors.

## 10.77 Output 77 Kaplan-Meier Curve of Overall Survival

Programming Note:

Analysis population: Safety
 Program name: G EF KM OS

# **Appendix 1 Region Categories**

We only display regions and countries here where actually patients were enrolled.

Input needed from Study SPA/BioStats: Add any other countries to this table if your study has a site there with patients enroled

| Region | Member Countries |
|-------------------|-------------------------------------------|
| Western Europe | Belgium, Finland, France, Germany, Italy, |
| | Spain, Sweden, United Kingdom |
| Eastern Europe | Czech Republic, Hungary, Russia |
| North America | Canada, United States |
| <mark>Asia</mark> | China, Japan, Taiwan, South Korea |
| Other | Australia, Israel, New Zealand |

# DAP M 2 Update Log

| Date | Section | Description | Author |
|---|---|---|---|
| 24MAY2017 | Output 57 | Changed Change from Baseline to Shift Table | |
| 16MAY2017 | Output36 | Added "Total number of patients with at least one AE" category instead of displaying sub-category under "Total number of patients with at least one" category | |
| 07JUN2017 | Output53 | Added "Other" as sub-category under "Causes of Death" category | |
| 14JUN2017 | Output5 | Updated "Induction Phase" categorie as "Induction started", similarly "Maintenance/Consolidation Phase" to "Maintenance/ Consolidation Phase started". Also added "Discontinued Induction" & "Discontinued Maintenance/Consolidation" categories. | |
| 17JUL2017 | Table<br>Selected AE | Removed tick for bo29561 for Late onset/prolonged neutropenia. Updated definition of Neutropenia for BO29561-3 | |
| 21JUL2017 | Table Selected AE/AESI Titles of summaries | Second Malignancy and TLS moved to AESI In Summaries titles 'Summary of' removed | |
| 26JUL2017 | Safety<br>Summary<br>(Ouput 36) | Removed last row as this is not part of original STREAM template and is not appropriate to use: No connection between related AE and AE given as reason for study discontinuation (based on study completion page) | |
| 08AUG2017 | Output 24 | Add programming note: Use visit instead of cycle for BO29561 and BO29563 | |
| 14AUG2017 | Table 6.2.2,<br>Title of AESI<br>outputs | AESI categories updated in Table. AESI renamed to 'potential AESI' in output titles. | |
| 11AUG2017 | 6.2.1, output<br>34, output<br>41 | In BO29561/2/3 additional AESI tables based on eCRF tickbox. | |
| 14Aug2017 | Output 78 | Use categories Low/Intermediate/High for FLIPI.<br>Low/High for IPI. | |
| 22AUG2017 | Table 6.2.2 | AESI category Hypersensitivity updated | |

| 17OCT2017 | 6.4.5 | Hy's law: use BL instead of ULN for AST/ALT |
|---|---|---|
| 29JAN2017 | output 36 | Added 2 rows into template |
| 06SEP2018 | Output53 | Removed "Deaths during the treatment are those occurred within 28 days after last study drug." footnote. |
| 100CT2018 | Table 6.2.2 | Added AESI category 'Auto-immune hemolytic anaemia', updated AESI categories for Diabetes mellitus and Rash as requested by email on 09OCT2018 |
| 17OCT2018 | Table 6.2.2 | Updated AESI categories IRR and myocarditis as requested by in email on 17OCT2018 |
| 10DEC2018 | 6.4.9 | Added HACA in this section |
| 29JAN2019 | 6.2.1/6.2.2 | Added conditions for Atezo specific AESI (onset >= cycle 2, causality to Atezo suspected) |